CLINICAL TRIAL: NCT01966445
Title: A Phase I, First Time in Human, Open-Label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Anti-Her3 Monoclonal Antibody GSK2849330 in Subjects With Advanced Her3-Positive Solid Tumors
Brief Title: Dose Escalation Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of GSK2849330 in Subjects With Advanced Her3-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117158; 2013-001699-39 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Cancer; Neoplasms
Keywords: GSK2849330; Oncology; First Time in Human; HER3
MeSH Terms: conditions — Neoplasms | interventions — GSK2849330

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2849330 Part 1 (Experimental): 1 hour infusion administered intravenously at intervals of one week or more (escalating doses).
  Interventions: Biological: GSK2849330
- GSK2849330 Part 2 (Experimental): Intravenous infusion administered at the dose and schedule established in Part 1
  Interventions: Biological: GSK2849330

INTERVENTIONS:
Biological: GSK2849330 — Solution containing 100 mg/millilter (mL) GSK2849330 for intravenous infusion

SUMMARY:
Human Epidermal Growth Factor Receptor 3 (HER3) expression is seen across a wide variety of solid malignancies and is associated with poor prognosis. Up-regulation of HER3 expression and activity is also associated with resistance to multiple pathway inhibitors. GSK2849330, a monoclonal antibody targeting HER3, is a new agent for subjects whose tumors express HER3. This study is a phase I, first time in human, open-label, dose escalation study. The purpose of this study is to investigate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of GSK2849330 in subjects with advanced HER3-positive solid tumors. The study will be conducted in two parts. Part 1 (Dose-Escalation Phase) will include dose escalation and PK/PD cohorts to evaluate safety, PK, and PD to guide selection of dose regimen(s) for Part 2. In Part 2 (Expansion Cohorts), up to 3 cohorts will be enrolled at the dose regimen(s) selected based on Part 1 data, to evaluate safety in a larger cohort of subjects at the recommended dose regimen and also to evaluate preliminary evidence of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >=18 years of age (at the time consent is obtained).
* Written informed consent provided.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Sufficient archival tumor specimen is available for HER3 immunohistochemistry (IHC) analysis, or subject is willing to undergo a fresh tumor biopsy for HER3 IHC analysis.
* Histologically or cytologically confirmed diagnosis of one of the following solid tumor malignancies for which no standard therapeutic alternatives exist: bladder cancer, breast cancer, castrate-resistant prostate cancer, cervical cancer, colorectal cancer (CRC), gastric cancer, hepatocellular carcinoma (HCC), melanoma, non-small cell lung cancer (NSCLC), ovarian cancer, pancreatic cancer, squamous cancers of the head and neck region (including parotid and nasopharynx).

Exclusion Criteria:

* Subjects with leptomeningeal or brain metastases or spinal cord compression.
* Prior HER3- directed treatment (HER2- or EGFR-directed treatment is acceptable).
* Concurrent medical condition that would jeopardize compliance.
* Receiving chronic immunosuppressive therapies (includes daily steroid doses in excess of 20 milligrams [mg]/day of prednisone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (10):
- United States (3):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (3):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam

REFERENCES:
- [Derived] Drilon A, Somwar R, Mangatt BP, Edgren H, Desmeules P, Ruusulehto A, Smith RS, Delasos L, Vojnic M, Plodkowski AJ, Sabari J, Ng K, Montecalvo J, Chang J, Tai H, Lockwood WW, Martinez V, Riely GJ, Rudin CM, Kris MG, Arcila ME, Matheny C, Benayed R, Rekhtman N, Ladanyi M, Ganji G. Response to ERBB3-Directed Targeted Therapy in NRG1-Rearranged Cancers. Cancer Discov. 2018 Jun;8(6):686-695. doi: 10.1158/2159-8290.CD-17-1004. Epub 2018 Apr 2. PMID 29610121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase 1 study of anti-human epidermal growth factor receptor 3 (HER3) antibody, GSK2849330 in participants with advanced solid tumors expressing HER3. The study was conducted in 2 parts-Part1 (dose escalation) and Part2 (dose expansion). The starting dose in Part1 was 1.4 milligrams per kilogram (mg/kg) GSK2849330 given weekly for 28 days
Pre-assignment Details: A total of 29 participants were randomized. The study was conducted in three countries. Participants in the GSK2849330 30 mg/kg weekly arm were not double counted with any other Arm.
Groups:
- Part1: GSK2849330 1.4 mg/kg Weekly: Participants were administered a weekly dose of 1.4 mg/kg GSK2849330 as intravenous infusion for 28 days
- Part1: GSK2849330 3 mg/kg Every 2 Weeks: Participants were administered 3 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days.
- Part1: GSK2849330 3 mg/kg Weekly: Participants were administered a weekly dose of 3 mg/kg GSK2849330 as intravenous infusion for 28 days.
- Part1: GSK2849330 10 mg/kg Every 2 Weeks: Participants were administered 10 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days.
- Part1: GSK2849330 30 mg/kg Every 2 Weeks: Participants were administered 30 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days
- Part1: GSK2849330 30 mg/kg Weekly; Part2: GSK2849330 30 mg/kg Weekly: Participants were administered a weekly dose of 30 mg/kg GSK2849330 as intravenous infusion for 28 days.
Period: Part1 (Median Exposure of 6.143 Weeks)
Arm/Group | Part1: GSK2849330 1.4 mg/kg Weekly | Part1: GSK2849330 3 mg/kg Every 2 Weeks | Part1: GSK2849330 3 mg/kg Weekly | Part1: GSK2849330 10 mg/kg Every 2 Weeks | Part1: GSK2849330 30 mg/kg Every 2 Weeks | Part1: GSK2849330 30 mg/kg Weekly | Part2: GSK2849330 30 mg/kg Weekly
Started | 1 | 3 | 2 | 5 | 4 | 5 | 0
Completed | 1 | 1 | 1 | 2 | 1 | 4 | 0
Not Completed | 0 | 2 | 1 | 3 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 2 | 0 | 0
Period: Part2 (Median Exposure of 7.143 Weeks)
Arm/Group | Part1: GSK2849330 1.4 mg/kg Weekly | Part1: GSK2849330 3 mg/kg Every 2 Weeks | Part1: GSK2849330 3 mg/kg Weekly | Part1: GSK2849330 10 mg/kg Every 2 Weeks | Part1: GSK2849330 30 mg/kg Every 2 Weeks | Part1: GSK2849330 30 mg/kg Weekly | Part2: GSK2849330 30 mg/kg Weekly
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Groups:
- GSK2849330 1.4 mg/kg Weekly: Participants were administered a weekly dose of 1.4 mg/kg GSK2849330 as intravenous infusion for 28 days
- GSK2849330 3 mg/kg Every 2 Weeks: Participants were administered 3 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days.
- GSK2849330 3 mg/kg Weekly: Participants were administered a weekly dose of 3 mg/kg GSK2849330 as intravenous infusion for 28 days.
- GSK2849330 10 mg/kg Every 2 Weeks: Participants were administered 10 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days.
- GSK2849330 30 mg/kg Every 2 Weeks: Participants were administered 30 mg/kg GSK2849330 as an intravenous infusion every 2 weeks for 28 days
- GSK2849330 30 mg/kg Weekly: Participants were administered a weekly dose of 30 mg/kg GSK2849330 as intravenous infusion for 28 days. The arm included participants receiving 30 mg/kg weekly from both Part 1 (dose-escalation cohort) and Part 2 (dose expansion cohort).
- Total: Total of all reporting groups
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly | Total
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (NA) — Standard deviation for 1.4 mg/kg weekly arm could not be calculated as only a single participant was analyzed in this arm. | 62.3 (4.04) | 46.0 (21.21) | 66.2 (7.19) | 58.3 (8.73) | 62.5 (11.65) | 61.4 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 2 | 2 | 5 | 13
  Male | 1 | 0 | 1 | 3 | 2 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Asian-Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race customized: White | 1 | 3 | 2 | 5 | 4 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Parts 1 and 2
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the outcomes mentioned; events of possible study treatment-induced liver injury with hyperbilirubinemia; and left ventricular ejection fraction (LVEF) meeting stopping criteria. AEs were collected in All Treated Population which comprised of all participants who received at least one dose of GSK2849330. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  AEs | 1 | 3 | 2 | 5 | 4 | 14
  SAEs | 0 | 1 | 0 | 1 | 1 | 3

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)-Parts 1 and 2
Description: An event was considered a DLT if it occured within the first 4 weeks (28 days) of treatment, and met one of the following criteria unless it could be established that the event was unrelated to treatment: Grade 3 or greater non-hematologic toxicity; Grade 4 neutropenia lasting >5 days; Febrile neutropenia, of any grade or duration; Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia associated with bleeding; Alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) with bilirubin >2 times ULN; Any Grade 2 or greater toxicity that in the judgment of the investigator and GlaxoSmithKline (GSK) Medical Monitor, would be considered dose-limiting; Grade 3 or greater decrease in LVEF. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Up to 28 days
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Parts 1 and 2
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (Total bil), calcium, creatinine, gamma glutamyl transferase (GGT), glucose, potassium, magnesium, sodium, phosphorus, uric acid. Laboratory parameters were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Baseline is the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Change from Baseline was calculated as visit value minus Baseline value. Data for worst-case post Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: All Treated Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Albumin; any Grade increase; n=1,3,2,5,4,14 | 1 | 1 | 0 | 3 | 3 | 6
  Albumin; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 1
  Albumin; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  ALP; any grade increase; n=1,3,2,5,4,14 | 1 | 0 | 1 | 1 | 1 | 7
  ALP; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 1 | 1
  ALP; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; any Grade increase; n=1,3,2,5,4,14 | 0 | 2 | 0 | 2 | 3 | 6
  ALT; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  ALT; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  AST; any Grade increase; n=1,3,2,5,4,14 | 0 | 1 | 0 | 2 | 2 | 5
  AST; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 1
  AST; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Total bil; any Grade increase; n=1,3,2,5,4,14 | 0 | 1 | 0 | 1 | 0 | 2
  Total bil; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Total bil; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium; any Grade increase; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 2 | 2
  Calcium; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 1 | 0
  Calcium; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; any Grade increase; n=1,3,2,5,4,14 | 0 | 1 | 0 | 1 | 1 | 2
  Creatinine; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  GGT; any Grade increase; n=1,3,2,5,4,14 | 1 | 0 | 1 | 2 | 3 | 8
  GGT; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 1 | 1 | 0 | 3
  GGT; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 1 | 0
  Glucose; any Grade increase; n=1,3,2,5,4,14 | 1 | 0 | 1 | 3 | 2 | 4
  Glucose; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium; any Grade increase; n=1,3,2,5,4,14 | 0 | 2 | 0 | 0 | 0 | 1
  Potassium; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium; any Grade increase; n=1,3,2,5,4,14 | 0 | 1 | 0 | 0 | 2 | 4
  Magnesium; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium; any Grade increase; n=1,3,2,5,4,14 | 0 | 1 | 0 | 0 | 3 | 4
  Sodium; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorus; any Grade increase; n=1,3,2,5,4,14 | 1 | 0 | 0 | 0 | 0 | 4
  Phosphorus; increase to Grade 3; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorus; increase to Grade 4; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 0
  Uric acid; any Grade increase; n=0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Uric acid; any Grade increase; n=0,0,0,0,0,1 |  |  |  |  |  | 1
  Uric acid; increase to Grade 3; n=0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Uric acid; increase to Grade 3; n=0,0,0,0,0,1 |  |  |  |  |  | 0
  Uric acid; increase to Grade 4; n=0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Uric acid; increase to Grade 4; n=0,0,0,0,0,1 |  |  |  |  |  | 1

4. Primary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry Data With Respect to Normal Range-Parts 1 and 2
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: direct bilirubin (D.Bil.), cancer antigen (CA)-125, CA-15.3, CA19-9, chloride, carbon dioxide (CO2)/bicarbonate (HCO3), luteinizing hormone (LH), total protein and urea or blood urea nitrogen (BUN). Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Change from Baseline was calculated as visit value minus Baseline value. A laboratory value that is outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Number of participants with change from Baseline in clinical chemistry data at worst-case post Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  D.Bil.; Decrease to Low; n=1,3,2,5,3,14: number analyzed (Participants) | 1 | 3 | 2 | 5 | 3 | 14
  D.Bil.; Decrease to Low; n=1,3,2,5,3,14 | 0 | 0 | 1 | 0 | 0 | 0
  D.Bil.; increase to high; n=1,3,2,5,3,14: number analyzed (Participants) | 1 | 3 | 2 | 5 | 3 | 14
  D.Bil.; increase to high; n=1,3,2,5,3,14 | 0 | 1 | 0 | 2 | 1 | 4
  CA-125; Decrease to Low; n=1,3,0,5,4, 0: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 0
  CA-125; Decrease to Low; n=1,3,0,5,4, 0 | 0 | 0 |  | 0 | 0 |
  CA-125; increase to high; n=1,3,0,5,4, 0: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 0
  CA-125; increase to high; n=1,3,0,5,4, 0 | 0 | 0 |  | 0 | 0 |
  CA 15.3; Decrease to Low; n=0, 0, 0, 0, 4, 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0
  CA 15.3; Decrease to Low; n=0, 0, 0, 0, 4, 0 |  |  |  |  | 0 |
  CA 15.3; increase to high; n=0, 0, 0, 0, 4, 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0
  CA 15.3; increase to high; n=0, 0, 0, 0, 4, 0 |  |  |  |  | 0 |
  CA 19-9.; Decrease to Low; n=1,0,0,0,2,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0
  CA 19-9.; Decrease to Low; n=1,0,0,0,2,0 | 0 |  |  |  | 0 |
  CA 19-9; increase to high; n=1,0,0,0,2,0: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0
  CA 19-9; increase to high; n=1,0,0,0,2,0 | 0 |  |  |  | 0 |
  Chloride; Decrease to Low; n=1,3,2,5,4,14 | 0 | 1 | 0 | 1 | 2 | 4
  Chloride; increase to high; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 0 | 1
  CO2/HCO3.; Decrease to Low; n=1,3,2,5,4,14 | 0 | 0 | 0 | 3 | 1 | 2
  CO2/HCO3; increase to high; n=1,3,2,5,4,14 | 0 | 1 | 0 | 1 | 0 | 7
  LH; Decrease to Low; n=1,0,2,3,2,7: number analyzed (Participants) | 1 | 0 | 2 | 3 | 2 | 7
  LH; Decrease to Low; n=1,0,2,3,2,7 | 0 |  | 0 | 0 | 0 | 1
  LH; increase to high; n=1,0,2,3,2,7: number analyzed (Participants) | 1 | 0 | 2 | 3 | 2 | 7
  LH; increase to high; n=1,0,2,3,2,7 | 0 |  | 0 | 0 | 0 | 3
  Total Protein; Decrease to Low; n=1,3,2,5,4,14 | 0 | 1 | 1 | 1 | 0 | 1
  Total Protein; increase to high; n=1,3,2,5,4,14 | 0 | 0 | 0 | 1 | 0 | 0
  Urea/BUN; Decrease to Low; n=1,3,2,5,4,14 | 0 | 0 | 0 | 0 | 1 | 3
  Urea/BUN; increase to high; n=1,3,2,5,4,14 | 0 | 1 | 1 | 0 | 0 | 2

5. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Parts 1 and 2
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, lymphocytes, total neutrophils, platelet count, and white blood cell (WBC). The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Change from Baseline was calculated as visit value minus Baseline value. Number of participants with any grade increase, increase to Grade 3 and increase to Grade 4 in hematology data at worst-case post Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Hemoglobin; any Grade increase | 0 | 1 | 0 | 0 | 3 | 7
  Hemoglobin; increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 2
  Hemoglobin; increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes; any grade increase | 0 | 0 | 1 | 3 | 1 | 5
  Lymphocytes; increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 2
  Lymphocytes; increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Total neutrophils; any Grade increase | 0 | 0 | 0 | 1 | 0 | 1
  Total neutrophils; increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Total neutrophils; increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet; any Grade increase | 0 | 1 | 1 | 0 | 0 | 0
  Platelet; increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet; increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  WBC; any Grade increase | 0 | 1 | 0 | 2 | 0 | 1
  WBC; increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  WBC; increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Change From Baseline in Hematology Data With Respect to Normal Range-Parts 1 and 2
Description: Blood samples were collected for the analysis of following hematology parameters: basophils, eosinophils, hematocrit, mean corpuscle hemoglobin concentration (MCHC), mean corpuscle hemoglobin (MCH), mean corpuscle volume (MCV), monocytes, red blood cell count (RBC) and reticulocytes. A laboratory value that was outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Change from Baseline was calculated as value at visit minus Baseline value. Number of participants with change from Baseline in hematology data at worst-case post Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Basophils: decrease to low | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: increase to high | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: decrease to low | 0 | 0 | 1 | 0 | 0 | 0
  Eosinophils: increase to high | 0 | 0 | 0 | 0 | 0 | 2
  Hematocrit: decrease to low | 0 | 0 | 0 | 1 | 1 | 4
  Hematocrit: increase to high | 0 | 0 | 0 | 0 | 0 | 0
  MCHC: decrease to low | 1 | 0 | 0 | 0 | 0 | 3
  MCHC: increase to high | 0 | 0 | 0 | 0 | 0 | 0
  MCH: decrease to low | 1 | 1 | 0 | 0 | 0 | 1
  MCH: increase to high | 0 | 0 | 0 | 0 | 1 | 0
  MCV: decrease to low | 0 | 1 | 0 | 0 | 0 | 1
  MCV: increase to high | 0 | 0 | 0 | 0 | 0 | 1
  Monocytes: decrease to low | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: increase to high | 1 | 0 | 0 | 0 | 0 | 2
  RBC: decrease to low | 0 | 0 | 0 | 3 | 0 | 7
  RBC: increase to high | 0 | 0 | 0 | 0 | 0 | 1
  Reticulocytes: decrease to low | 0 | 0 | 0 | 1 | 0 | 2
  Reticulocytes: increase to high | 0 | 0 | 0 | 1 | 2 | 3

7. Primary Outcome: Number of Participants With Change From Baseline in Urinalysis Data With Respect to Normal Range-Parts 1 and 2
Description: Urine samples were collected for the analysis of urine potential of hydrogen (pH) and urine specific gravity. A laboratory value that was outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date. Change from Baseline was calculated as visit value minus Baseline value. The data for worst-case post Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Urine pH; decrease to low; n=1, 3, 1, 5, 4, 7: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 7
  Urine pH; decrease to low; n=1, 3, 1, 5, 4, 7 | 0 | 0 | 0 | 0 | 0 | 0
  Urine pH; increase to high; n=1, 3, 1, 5, 4, 7: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 7
  Urine pH; increase to high; n=1, 3, 1, 5, 4, 7 | 0 | 0 | 0 | 0 | 0 | 1
  Specific gravity; decrease to low; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  Specific gravity; decrease to low; n=1,3,1,4,4,8 | 0 | 1 | 0 | 0 | 0 | 0
  Specific gravity; increase to high; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  Specific gravity; increase to high; n=1,3,1,4,4,8 | 1 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Change From Baseline in Vital Signs-Parts 1 and 2
Description: Vital sign measurements included systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature (Temp) and heart rate (HR). Vital signs were graded according to NCI-CTCAE version 4.0. The following criteria was used to flag vital signs of potential clinical importance: change from Baseline in HR (decrease to <60 beats per minute and increase to >100 beats per minute); increase in SBP from Baseline (>=120 to <140 millimeters of mercury [mmHg] Grade 1; >=140 to <160 mmHg [Grade 2]; >=160 [Grade 3]); increase in DBP from Baseline (>=80 to <90 [Grade 1]; >=90 to <100 [Grade 2]; >=100 mmHg [Grade 3]) and change in temperature from Baseline (increase to >=38 or decrease to <=35 degree Centigrade). Baseline was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was calculated as visit value minus Baseline value. The data for worst-case post Baseline is presented.
Time Frame: Baseline and median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  HR; decrease to <60 beats per minute | 1 | 1 | 0 | 2 | 0 | 4
  HR; increase to >100 beats per minute | 0 | 0 | 1 | 1 | 0 | 5
  Temp; decrease to <=35 degree Celsius | 0 | 0 | 0 | 1 | 0 | 0
  Temp; increase to >=38 degree Celsius | 0 | 0 | 0 | 0 | 0 | 4
  SBP; increase to Grade 1 (120-139 mmHg) | 0 | 0 | 2 | 1 | 2 | 3
  SBP; increase to Grade 2 (140-159 mmHg) | 0 | 0 | 0 | 1 | 0 | 4
  SBP; increase to Grade 3 (>=160 mmHg) | 0 | 1 | 0 | 1 | 2 | 0
  DBP; increase to Grade 1 (80-89 mmHg) | 0 | 1 | 2 | 3 | 1 | 7
  DBP; increase to Grade 2 (90-99 mmHg) | 0 | 1 | 0 | 0 | 0 | 1
  DBP; increase to Grade 3 (>=100 mmHg) | 0 | 0 | 0 | 1 | 0 | 1

9. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings-Parts 1 and 2
Description: A 12-lead ECG was measured using an automated ECG machine after at least 5 minutes of rest for the participant in a semi-recumbent or supine position. Number of participants with abnormal ECG findings at any time post-Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Abnormal-not clinically significant | 1 | 3 | 1 | 4 | 3 | 4
  Abnormal-clinically significant | 0 | 0 | 0 | 0 | 0 | 1

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK2849330-Part 1
Description: The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data is defined as Cmax. Blood samples were collected at indicated time points. The analysis was performed on pharmacokinetic (PK) parameter population which comprised of all participants from the PK concentration population (participants who received at least one dose of GSK2849330 and for whom at least one post-dose PK sample was obtained and analyzed) for whom valid and valuable PK parameters were derived.
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- GSK2849330 30 mg/kg Weekly: Participants were administered a weekly dose of 30 mg/kg GSK2849330 as intravenous infusion for 28 days. The arm included participants receiving 30 mg/kg weekly from Part 1 (dose-escalation cohort).
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 3 | 5
Nanograms per milliliter | 29790.0 (NA) — The geometric coefficient of variation could not be calculated as a single participant was analyzed at the specified time point. | 62495.2 (34.8) | 83845.0 (24.1) | 233997.8 (2.7) | 639127.3 (45.4) | 778470.6 (14.5)

11. Secondary Outcome: Cmax of GSK2849330-Part 2
Description: PK parameters for Part 2 were not analyzed due to sparse sampling. The protocol was written in a flexible way to either pursue or not pursue additional analyses in Part 2.
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population. PK parameters for Part 2 were not analyzed due to sparse sampling.
Groups:
- GSK2849330 30 mg/kg Weekly: Participants were administered a weekly dose of 30 mg/kg GSK2849330 as intravenous infusion for 28 days. The arm included participants receiving 30 mg/kg weekly in Part 2 (dose expansion cohort).
Arm/Group | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 0

12. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for GSK2849330-Part 1
Description: The time at which Cmax is observed was determined directly from the raw concentration-time data is defined as Tmax. Blood samples were collected at indicated time points for evaluation of pharmacokinetic parameters.
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 3 | 5
Hours | 2.070 [2.070 to 2.070] | 2.130 [2.000 to 6.170] | 88.035 [6.370 to 169.700] | 2.280 [2.130 to 6.000] | 3.280 [2.300 to 6.230] | 2.100 [1.830 to 2.330]

13. Secondary Outcome: Tmax for GSK2849330-Part 2
Description: as for outcome 11
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population. PK parameters for Part 2 were not analyzed due to sparse sampling.
Arm/Group | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 0

14. Secondary Outcome: Area Under the Concentration Time Curve (AUC) to a Fixed Nominal Time (AUC[0 to 168]) and AUC(0 to 336) for GSK2849330-Part 1
Description: The AUC to a fixed nominal time AUC(0-168) and AUC(0-336) were calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples were collected at indicated time points for determination of PK parameters.
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 3 | 5
Hours*nanogram per milliliter
  AUC(0 to 168); n=1, 3, 2, 3, 3, 5 | 1962762.0 (NA) — Geometric coefficient of variation could not be calculated as a single participant was analyzed at the specified time point. | 5787797.8 (27.2) | 618552.6 (20559.2) | 18185733.6 (28.8) | 54346531.5 (30.2) | 54388333.7 (22.6)
  AUC(0 to 336); 0, 3, 0, 3, 3, 0: number analyzed (Participants) | 0 | 3 | 0 | 3 | 3 | 0
  AUC(0 to 336); 0, 3, 0, 3, 3, 0 |  | 7855808.8 (28.7) |  | 23409694.6 (39.4) | 72404738.6 (34.2) |

15. Secondary Outcome: AUC(0 to 168) and AUC(0 to 336) for GSK2849330-Part 2
Description: as for outcome 11
Time Frame: Day 1 (pre-dose, 1 and 6 hours post-dose), Day 8, Day 15, Day 29, and every 12 weeks from first dose
Population: PK Parameter Population. PK parameters for Part 2 were not analyzed due to sparse sampling.
Arm/Group | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 0

16. Secondary Outcome: Serum HER3 From Tumor Tissue-Parts 1 and 2
Description: Pre-treatment and on-treatment biopsy tissues (tumor and normal skin) were analyzed for markers of HER3 pathway such as HER3 that may indicate a pharmacodynamic (PD) response to GSK2849330. Serum HER3 (soluble HER3) analyses was performed. The analysis was performed on PD population which comprised of all participants who received at least one dose of GSK2849330 and for whom at least one evaluable paired pre-treatment PD sample and on-treatment PD sample were obtained and analyzed. Mean and standard deviation for serum HER3 is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Day 1 (pre-dose, 1 hour, 6 hours), Day 2, Day 8, Day 15, Day 29 and follow-up (28 days post last dose)
Population: PD Population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanomoles
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 12
Nanomoles
  Day 1; pre-dose; n=1, 3, 1, 5, 4, 12 | 13.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.11 (2.603) | 16.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.42 (4.004) | 13.67 (4.681) | 11.08 (5.322)
  Day 1; 1 hour; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  Day 1; 1 hour; n=1, 3, 1, 5, 4, 11 | 11.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.14 (2.966) | 7.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.76 (2.228) | 9.55 (4.437) | 5.59 (2.709)
  Day 1; 6 hours; n=1, 3, 1, 5, 4, 10: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 10
  Day 1; 6 hours; n=1, 3, 1, 5, 4, 10 | 9.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.71 (2.679) | 12.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.69 (4.058) | 9.39 (4.586) | 5.35 (2.031)
  Day 2; n=0, 0, 1, 1, 1, 2: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 2
  Day 2; n=0, 0, 1, 1, 1, 2 |  |  | 8.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 3.50 (2.001)
  Day 8; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  Day 8; n=1, 3, 1, 5, 4, 11 | 10.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.59 (4.353) | 10.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.85 (3.771) | 6.32 (2.702) | 6.05 (2.382)
  Day 15; n=0, 2, 1, 3, 4, 10: number analyzed (Participants) | 0 | 2 | 1 | 3 | 4 | 10
  Day 15; n=0, 2, 1, 3, 4, 10 |  | 10.62 (1.110) | 7.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.38 (3.535) | 9.84 (3.127) | 4.66 (1.402)
  Day 29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  Day 29; n=1, 3, 1, 4, 4, 8 | 10.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.18 (3.695) | 7.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.60 (3.220) | 6.91 (4.621) | 4.13 (1.815)
  Follow-up; n=1, 2, 1, 3, 2, 5: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 5
  Follow-up; n=1, 2, 1, 3, 2, 5 | 6.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.22 (3.090) | 14.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.41 (1.406) | 3.73 (0.424) | 4.39 (2.975)

17. Secondary Outcome: Overall Response Rate (ORR)-Parts 1 and 2
Description: ORR was determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST v 1.1). ORR was calculated as the number of participants with best overall response of complete response (CR) and partial response (PR). CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in the short axis and PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters (e.g., percent change from Baseline). An estimate to the true response rate for the number of participants analyzed is given. The 95% confidence interval was the exact confidence interval based on binomial proportion for ORR. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Median of 6.143 weeks of drug exposure
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants | 0 [0.0 to 97.5] | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 1 [0.2 to 33.9]

18. Secondary Outcome: Number of Participants With Antibodies to GSK2849330 in Serum
Description: Serum samples were collected for the determination of anti-GSK2849330 antibodies using a validated immunoelectrochemiluminescent (ECL) assay. The assay involved screening, confirmation and titration steps (tiered-testing approach). If serum samples contained anti-GSK2849330 antibodies, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. The number of participants who tested positive for anti-GSK2849330 antibody in confirmatory testing on Day 1 and at any time post-Baseline is presented. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Median of 6.143 weeks of drug exposure
Population: All Treated Population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 14
Participants
  Day1; n=1, 3, 2, 5, 4, 13: number analyzed (Participants) | 1 | 3 | 2 | 5 | 4 | 13
  Day1; n=1, 3, 2, 5, 4, 13 | 0 | 0 | 0 | 0 | 0 | 1
  Any time post-Baseline; n=1, 3, 1, 5, 4, 7: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 7
  Any time post-Baseline; n=1, 3, 1, 5, 4, 7 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Cluster of Differentiation (CD) Marker
Description: Blood samples were collected on Day (D) 1 at pre-dose (pre) and at 1 hour (h) and 6 h post infusion for the analysis of markers to evaluate biological activity of GSK2849330. A pre-dose blood sample was collected on D8, D15 and D29 with additional blood sample collected at progression of disease. CDX241 represent CD45+CD3-CD56+CD16+CD69+CD107+, CDX243=CD45+CD3-CD56+CD16+CD69+CD107-; CDX244=CD45+CD3-CD56+CD16+CD69-CD107+ and CDX245=CD45+CD3-CD56+CD16+CD69-CD107-. For participants in GSK2849330 3 mg/kg weekly arm, two samples (S1 and S2) were collected for D15 analysis. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Time Frame: Median of 6.143 weeks of drug exposure
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percentage of CD marker cells
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
Number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 12
Percentage of CD marker cells
  CD45+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+; D1; pre; n=1, 3, 1, 5, 4, 9 | 99.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.83 (0.058) | 99.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.76 (0.434) | 99.93 (0.050) | 101.57 (6.268)
  CD45+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 99.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.87 (0.058) | 99.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.76 (0.434) | 99.93 (0.050) | 101.13 (4.656)
  CD45+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 99.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.83 (0.058) | 99.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.8 (0.255) | 99.93 (0.096) | 101.02 (3.978)
  CD45+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 99.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.7 (0.424) |  | 99.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+; D8; n=1, 3, 0, 5, 4, 8 | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.87 (0.058) |  | 99.4 (1.231) | 99.80 (0.400) | 99.75 (0.576)
  CD45+; D15;S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+; D15;S1; n=1, 3, 1, 5, 4, 9 | 99.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.90 (0.000) | 99.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.78 (0.327) | 99.78 (0.320) | 100.33 (2.495)
  CD45+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+; D15; S2; n=0,0,1,0,0,0 |  |  | 99.8 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+; D29; n=1, 3, 1, 4, 4, 8 | 99.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.93 (0.058) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.78 (0.222) | 99.75 (0.436) | 100.80 (3.746)
  CD45+; follow-up (FU); n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+; follow-up (FU); n=1, 2, 0, 3, 1, 4 | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.85 (0.071) |  | 99.63 (0.551) | 99.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 101.60 (4.827)
  CD45+; unscheduled (USC); n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+; unscheduled (USC); n=0, 0, 1, 0, 0, 0 |  |  | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+; D1; pre;n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+; D1; pre;n=1, 3, 1, 5, 4, 9 | 62.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.00 (13.313) | 58.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 86.88 (2.580) | 71.98 (10.832) | 72.91 (8.027)
  CD45+CD3+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 76.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 73.83 (9.646) | 57.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 87.08 (2.153) | 75.80 (6.933) | 74.36 (9.552)
  CD45+CD3+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 81.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.43 (12.784) | 62.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 86.88 (2.580) | 77.83 (5.065) | 72.16 (10.282)
  CD45+CD3+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 48.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 86.60 (0.566) |  | 77.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+; D8; n=1, 3, 0, 5, 4, 8 | 72.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.67 (17.310) |  | 86.30 (1.505) | 77.53 (7.566) | 75.31 (8.234)
  CD45+CD3+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+; D15; S1; n=1, 3, 1, 5, 4, 9 | 73.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.97 (19.410) | 36.8 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 87.52 (1.359) | 76.08 (8.844) | 76.50 (5.723)
  CD45+CD3+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+; D15; S2; n=0,0,1,0,0,0 |  |  | 48.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+; D29; n=1, 3, 1, 4, 4, 8 | 76.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.97 (17.609) | 36.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 87.30 (1.753) | 73.58 (9.783) | 74.49 (12.798)
  CD45+CD3+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+; FU; n=1, 2, 0, 3, 1, 4 | 64.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.15 (7.425) |  | 83.53 (7.966) | 42.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.13 (11.425)
  CD45+CD3+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 58.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+; D1; pre;n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+; D1; pre;n=1, 3, 1, 5, 4, 9 | 9.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.67 (6.929) | 21.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.14 (22.721) | 24.95 (13.644) | 25.39 (11.076)
  CD45+CD3+CD8+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 8.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.20 (3.538) | 20.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.24 (21.617) | 20.48 (10.935) | 23.18 (10.434)
  CD45+CD3+CD8+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 8.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.47 (2.548) | 23.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 30.82 (22.379) | 23.38 (11.738) | 22.86 (11.701)
  CD45+CD3+CD8+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 21.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.70 (7.071) |  | 40.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+; D8; n=1, 3, 0, 5, 4, 8 | 10.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.70 (4.987) |  | 35.24 (22.320) | 24.60 (12.511) | 23.76 (9.382)
  CD45+CD3+CD8+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+; D15; S1; n=1, 3, 1, 5, 4, 9 | 9.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.90 (6.843) | 13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 36.46 (22.405) | 26.25 (13.843) | 27.00 (11.668)
  CD45+CD3+CD8+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+; D15; S2; n=0,0,1,0,0,0 |  |  | 15.7 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+; D29; n=1, 3, 1, 4, 4, 8 | 11.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.93 (6.110) | 17.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 40.85 (23.034) | 23.05 (11.997) | 20.40 (13.234)
  CD45+CD3+CD8+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+; FU; n=1, 2, 0, 3, 1, 4 | 7.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.55 (4.455) |  | 45.10 (29.487) | 6.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.88 (4.661)
  CD45+CD3+CD8+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 21.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-; D1; pre n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-; D1; pre n=1, 3, 1, 5, 4, 9 | 50.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 45.90 (9.124) | 36.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.76 (20.204) | 45.58 (4.365) | 47.71 (14.059)
  CD45+CD3+CD8-; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 66.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.77 (8.732) | 36.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 54.92 (19.213) | 53.90 (6.349) | 51.10 (17.633)
  CD45+CD3+CD8-; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 72.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 54.10 (13.421) | 36.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.26 (19.752) | 53.28 (10.943) | 49.26 (17.654)
  CD45+CD3+CD8-; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-; D2; n=0, 0, 1, 2, 0, 1 |  |  | 26.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 66.35 (7.425) |  | 36.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-; D8; n=1, 3, 0, 5, 4, 8 | 63.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 46.80 (12.759) |  | 50.48 (21.133) | 51.70 (11.040) | 51.48 (8.065)
  CD45+CD3+CD8-; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-; D15; S1; n=1, 3, 1, 5, 4, 9 | 63.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 48.37 (12.659) | 24.3 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.56 (21.357) | 49.60 (9.910) | 49.08 (13.029)
  CD45+CD3+CD8-; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-; D15; S2; n=0,0,1,0,0,0 |  |  | 36.1 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-; D29; n=1, 3, 1, 4, 4, 8 | 65.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 49.10 (12.137) | 19.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 45.55 (21.821) | 50.43 (3.402) | 54.63 (13.806)
  CD45+CD3+CD8-; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-; FU; n=1, 2, 0, 3, 1, 4 | 56.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.50 (3.394) |  | 38.20 (21.565) | 36.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 37.53 (16.020)
  CD45+CD3+CD8-; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-; USC; n=0, 0, 1, 0, 0, 0 |  |  | 38.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+; D1; pre n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+; D1; pre n=1, 3, 1, 5, 4, 9 | 24.3 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.50 (7.375) | 25.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.96 (1.757) | 13.83 (12.467) | 10.63 (8.253)
  CD45+CD3-CD16+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 9.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.03 (5.972) | 32.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.44 (2.411) | 8.00 (8.198) | 8.90 (6.203)
  CD45+CD3-CD16+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 3.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.80 (6.538) | 23.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 3.30 (2.314) | 6.43 (4.407) | 7.44 (4.569)
  CD45+CD3-CD16+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 35.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 2.50 (0.566) |  | 4.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+; D8; n=1, 3, 0, 5, 4, 8 | 11.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.71 (12.293) |  | 5.62 (3.128) | 9.23 (5.762) | 11.23 (7.852)
  CD45+CD3-CD16+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+; D15; S1; n=1, 3, 1, 5, 4, 9 | 11.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.73 (11.816) | 47.7 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.54 (3.138) | 9.50 (6.470) | 10.33 (7.555)
  CD45+CD3-CD16+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+; D15; S2; n=0,0,1,0,0,0 |  |  | 7.6 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+; D29; n=1, 3, 1, 4, 4, 8 | 11.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.83 (9.530) | 37.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.75 (2.654) | 10.73 (9.999) | 11.93 (7.323)
  CD45+CD3-CD16+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+; FU; n=1, 2, 0, 3, 1, 4 | 20.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.65 (4.031) |  | 6.67 (2.237) | 43.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.03 (10.920)
  CD45+CD3-CD16+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 19.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+; D1; pre; n=1, 3, 1, 5, 4, 9 | 25.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.03 (5.636) | 25.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.88 (1.221) | 15.93 (11.588) | 12.16 (7.479)
  CD45+CD3-CD56+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 10.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.13 (4.562) | 32.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.30 (1.581) | 10.50 (7.470) | 10.74 (6.300)
  CD45+CD3-CD56+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 4.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.47 (5.934) | 26.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.70 (1.913) | 9.43 (3.079) | 10.71 (7.319)
  CD45+CD3-CD56+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 42.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.10 (0.141) |  | 5.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+; D8; n=1, 3, 0, 5, 4, 8 | 13.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.43 (10.625) |  | 6.16 (2.574) | 11.10 (4.808) | 12.33 (7.733)
  CD45+CD3-CD56+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+; D15; S1; n=1, 3, 1, 5, 4, 9 | 13.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.53 (11.288) | 50.2 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.96 (2.266) | 11.73 (6.548) | 8.39 (4.622)
  CD45+CD3-CD56+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+; D15; S2; n=0,0,1,0,0,0 |  |  | 8.7 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+; D29; n=1, 3, 1, 4, 4, 8 | 13.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.90 (8.502) | 42.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.18 (2.428) | 13.73 (9.582) | 12.48 (9.517)
  CD45+CD3-CD56+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+; FU; n=1, 2, 0, 3, 1, 4 | 22.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.80 (1.556) |  | 8.37 (3.493) | 44.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.95 (8.912)
  CD45+CD3-CD56+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 22.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+; D1; pre; n=1, 3, 1, 5, 4, 9 | 3.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.17 (8.905) | 2.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.18 (10.303) | 6.20 (4.774) | 4.67 (2.707)
  CD45+CD3+CD56+; D1; 1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+; D1; 1 h; n=1, 3, 1, 5, 4, 9 | 1.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.03 (8.410) | 1.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.70 (7.601) | 6.65 (7.102) | 4.20 (3.321)
  CD45+CD3+CD56+; D1; 6 h; n=1, 3, 1, 5, 4, 11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+; D1; 6 h; n=1, 3, 1, 5, 4, 11 | 1.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.87 (7.566) | 13.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.50 (11.924) | 8.50 (10.745) | 4.17 (3.299)
  CD45+CD3+CD56+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 3.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.90 (14.001) |  | 7.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+; D8; n=1, 3, 0, 5, 4, 8 | 3.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.23 (8.977) |  | 12.36 (8.813) | 5.83 (2.756) | 3.49 (2.801)
  CD45+CD3+CD56+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+; D15; S1; n=1, 3, 1, 5, 4, 9 | 2.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.40 (8.118) | 1.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.48 (12.640) | 8.15 (3.746) | 4.43 (3.015)
  CD45+CD3+CD56+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+; D15; S2; n=0,0,1,0,0,0 |  |  | 1.3 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+; D29; n=1, 3, 1, 4, 4, 8 | 2.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.33 (8.629) | 3.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.88 (5.197) | 11.78 (9.751) | 2.91 (2.635)
  CD45+CD3+CD56+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+; FU; n=1, 2, 0, 3, 1, 4 | 2.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.20 (13.294) |  | 16.07 (6.757) | 3.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.10 (2.665)
  CD45+CD3+CD56+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 1.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD56+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD56+; D1; pre; n=1, 3, 1, 5, 4, 9 | 23.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.23 (6.307) | 23.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.48 (1.638) | 13.25 (12.307) | 9.58 (7.480)
  CD45+CD3-CD16+CD56+; D1;1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD56+; D1;1 h; n=1, 3, 1, 5, 4, 9 | 9.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.10 (5.237) | 31.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 3.98 (2.244) | 7.65 (8.118) | 7.98 (5.768)
  CD45+CD3-CD16+CD56+; D1;6 h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD56+; D1;6 h; n=1,3,1,5,4,11 | 3.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.90 (5.403) | 19.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 2.92 (2.348) | 6.10 (4.221) | 6.22 (4.445)
  CD45+CD3-CD16+CD56+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD56+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 33.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 2.40 (0.566) |  | 4.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD56+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD56+; D8; n=1, 3, 0, 5, 4, 8 | 10.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.33 (10.979) |  | 5.00 (2.891) | 8.68 (5.465) | 8.96 (6.217)
  CD45+CD3-CD16+CD56+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD56+; D15; S1; n=1, 3, 1, 5, 4, 9 | 10.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.93 (11.007) | 43.5 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.14 (2.926) | 8.88 (6.357) | 6.54 (4.360)
  CD45+CD3-CD16+CD56+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD56+; D15; S2; n=0,0,1,0,0,0 |  |  | 5.4 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD56+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD56+; D29; n=1, 3, 1, 4, 4, 8 | 10.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.20 (8.542) | 32.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.05 (2.357) | 10.18 (9.932) | 9.30 (6.776)
  CD45+CD3-CD16+CD56+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD56+; FU; n=1, 2, 0, 3, 1, 4 | 19.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.50 (3.111) |  | 6.07 (2.566) | 41.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.20 (9.937)
  CD45+CD3-CD16+CD56+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD56+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 18.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD19+; D1; pre n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+; D1; pre n=1, 3, 1, 5, 4, 9 | 9.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.67 (4.936) | 12.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.36 (3.364) | 9.48 (4.769) | 8.39 (3.194)
  CD45+CD3-CD19+; D1;1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+; D1;1 h; n=1, 3, 1, 5, 4, 9 | 11.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.77 (3.323) | 8.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.04 (3.492) | 11.53 (6.211) | 9.18 (3.819)
  CD45+CD3-CD19+; D1;6 h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD19+; D1;6 h; n=1,3,1,5,4,11 | 11.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.23 (3.329) | 6.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.36 (3.817) | 10.83 (6.636) | 9.00 (4.988)
  CD45+CD3-CD19+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD19+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 6.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.10 (0.141) |  | 10.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD19+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD19+; D8; n=1, 3, 0, 5, 4, 8 | 10.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.77 (4.701) |  | 5.76 (3.895) | 9.63 (4.786) | 7.65 (4.176)
  CD45+CD3-CD19+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+; D15; S1; n=1, 3, 1, 5, 4, 9 | 10.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.03 (6.116) | 7.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.10 (3.180) | 9.25 (4.339) | 8.90 (4.170)
  CD45+CD3-CD19+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD19+; D15; S2; n=0,0,1,0,0,0 |  |  | 26.2 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD19+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD19+; D29; n=1, 3, 1, 4, 4, 8 | 8.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.37 (7.392) | 13.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.10 (3.995) | 10.53 (6.106) | 7.44 (4.324)
  CD45+CD3-CD19+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD19+; FU; n=1, 2, 0, 3, 1, 4 | 10.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.05 (4.313) |  | 6.17 (8.361) | 8.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.33 (6.019)
  CD45+CD3-CD19+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD19+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 15.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD14+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+; D1; pre; n=1, 3, 1, 5, 4, 9 | 5.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.87 (0.971) | 10.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.58 (1.293) | 7.15 (2.029) | 4.87 (1.406)
  CD45+CD14+; D1;1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+; D1;1 h; n=1, 3, 1, 5, 4, 9 | 1.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 3.63 (2.103) | 11.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.20 (1.461) | 4.68 (2.926) | 3.52 (1.713)
  CD45+CD14+; D1;6 h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD14+; D1;6 h; n=1,3,1,5,4,11 | 4.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.37 (2.804) | 11.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.24 (1.756) | 5.80 (2.389) | 5.23 (2.581)
  CD45+CD14+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD14+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 5.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.10 (2.828) |  | 4.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD14+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD14+; D8; n=1, 3, 0, 5, 4, 8 | 7.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.30 (0.872) |  | 6.60 (1.594) | 7.10 (2.223) | 5.40 (2.115)
  CD45+CD14+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+; D15; S1; n=1, 3, 1, 5, 4, 9 | 4.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.60 (1.652) | 5.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.66 (1.108) | 6.93 (1.823) | 5.47 (3.061)
  CD45+CD14+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD14+; D15; S2; n=0,0,1,0,0,0 |  |  | 18.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD14+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD14+; D29; n=1, 3, 1, 4, 4, 8 | 5.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.93 (0.231) | 7.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.53 (1.162) | 6.68 (2.241) | 4.61 (1.108)
  CD45+CD14+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD14+; FU; n=1, 2, 0, 3, 1, 4 | 7.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.50 (1.273) |  | 8.03 (0.862) | 2.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.98 (1.692)
  CD45+CD14+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD14+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 8.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+; D1; pre; n=1, 3, 1, 5, 4, 9 | 67.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.37 (3.710) | 83.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.92 (7.038) | 82.50 (3.378) | 75.71 (15.845)
  CD45+CD3-CD16+CD69+; D1;1 h; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+; D1;1 h; n=1, 3, 1, 5, 4, 9 | 76.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.76 (2.213) | 87.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 81.88 (8.557) | 86.01 (3.898) | 78.53 (16.993)
  CD45+CD3-CD16+CD69+; D1;6 h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD69+; D1;6 h; n=1,3,1,5,4,11 | 77.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.99 (12.536) | 90.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 84.25 (5.802) | 84.57 (4.448) | 79.79 (12.178)
  CD45+CD3-CD16+CD69+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD69+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 91.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 89.03 (3.776) |  | 88.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD69+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD69+; D8; n=1, 3, 0, 5, 4, 8 | 77.29 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 75.83 (5.870) |  | 81.34 (10.373) | 79.91 (2.014) | 70.93 (21.532)
  CD45+CD3-CD16+CD69+; D15;S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+; D15;S1; n=1, 3, 1, 5, 4, 9 | 81.61 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.04 (3.286) | 96.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.28 (6.867) | 81.68 (7.216) | 78.53 (20.178)
  CD45+CD3-CD16+CD69+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+; D15;S2; n=0,0,1,0,0,0 |  |  | 92.76 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD69+; D29; n=1, 3, 1, 4, 4, 8 | 79.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 81.92 (2.273) | 85.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.73 (6.688) | 83.00 (6.240) | 74.56 (17.788)
  CD45+CD3-CD16+CD69+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD69+; FU; n=1, 2, 0, 3, 1, 4 | 77.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 84.40 (1.506) |  | 81.52 (12.737) | 76.46 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.85 (19.555)
  CD45+CD3-CD16+CD69+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 64.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD107+; D1; pre; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD107+; D1; pre; n=1, 3, 1, 5, 4, 9 | 7.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.40 (5.851) | 18.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.27 (13.221) | 23.96 (12.309) | 25.04 (30.481)
  CD45+CD3-CD16+CD107+; D1;1 h; n=1, 3, 1, 5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD107+; D1;1 h; n=1, 3, 1, 5,4,9 | 12.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.18 (8.160) | 8.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.43 (13.416) | 24.66 (13.827) | 23.16 (24.866)
  CD45+CD3-CD16+CD107+; D1;6 h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD107+; D1;6 h; n=1,3,1,5,4,11 | 14.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.30 (6.477) | 40.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 32.01 (16.156) | 21.55 (12.001) | 21.82 (17.204)
  CD45+CD3-CD16+CD107+; D2; n=0, 0, 1, 2, 0, 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD107+; D2; n=0, 0, 1, 2, 0, 1 |  |  | 26.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.96 (9.454) |  | 30.82 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD107+; D8; n=1, 3, 0, 5, 4, 8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD107+; D8; n=1, 3, 0, 5, 4, 8 | 33.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.90 (3.044) |  | 22.42 (10.572) | 14.43 (1.615) | 27.85 (27.884)
  CD45+CD3-CD16+CD107+; D15; S1; n=1, 3, 1, 5, 4, 9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD107+; D15; S1; n=1, 3, 1, 5, 4, 9 | 17.29 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.72 (4.937) | 38.6 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.00 (8.663) | 18.30 (3.558) | 21.68 (15.816)
  CD45+CD3-CD16+CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 65.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD107+; D29; n=1, 3, 1, 4, 4, 8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD107+; D29; n=1, 3, 1, 4, 4, 8 | 16.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.78 (3.719) | 52.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.08 (4.869) | 27.70 (12.686) | 17.22 (6.799)
  CD45+CD3-CD16+CD107+; FU; n=1, 2, 0, 3, 1, 4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD107+; FU; n=1, 2, 0, 3, 1, 4 | 14.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.49 (13.902) |  | 31.28 (29.410) | 11.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.42 (15.633)
  CD45+CD3-CD16+CD107+; USC; n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD107+; USC; n=0, 0, 1, 0, 0, 0 |  |  | 16.51 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+CD107+; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107+; D1; pre; n=1,3,1,5,4,9 | 6.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.33 (5.869) | 18.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.05 (12.990) | 23.53 (11.967) | 24.68 (30.659)
  CD45+CD3-CD16+CD69+CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107+; D1;1 h;n=1,3,1,5,4,9 | 11.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.86 (7.795) | 8.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.29 (13.208) | 24.42 (13.709) | 22.85 (24.965)
  CD45+CD3-CD16+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 14.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.29 (6.364) | 38.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.96 (16.199) | 21.33 (11.655) | 21.34 (17.411)
  CD45+CD3-CD16+CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 26.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.42 (10.218) |  | 30.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD69+CD107+; D8; n=1,3,0,5,4,8 | 32.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.77 (3.013) |  | 22.35 (10.534) | 14.40 (1.591) | 27.19 (27.949)
  CD45+CD3-CD16+CD69+CD107+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107+; D15; S1;n=1,3,1,5,4,9 | 16.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.60 (4.890) | 38.6 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.94 (8.669) | 18.11 (3.584) | 21.11 (16.206)
  CD45+CD3-CD16+CD69+CD107+; D15; S2;n=0,0,1,0,0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+CD107+; D15; S2;n=0,0,1,0,0, 0 |  |  | 64.8 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD69+CD107+; D29; n=1,3,1,4,4,8 | 16.42 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.70 (3.598) | 50.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.76 (4.922) | 27.36 (12.492) | 16.08 (6.127)
  CD45+CD3-CD16+CD69+CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD69+CD107+; FU; n=1,2,0,3,1,4 | 14.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.24 (13.548) |  | 31.06 (29.550) | 11.56 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.16 (15.866)
  CD45+CD3-CD16+CD69+CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+CD107+; USC; n=0,0,1,0,0,0 |  |  | 15.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+CD107-; D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107-; D1;pre; n=1,3,1,5,4,9 | 61.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.04 (7.996) | 65.29 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.87 (9.438) | 58.97 (12.115) | 51.03 (22.210)
  CD45+CD3-CD16+CD69+CD107-; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107-; D1;1 h;n=1,3,1,5,4,9 | 65.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.90 (8.250) | 78.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.59 (8.489) | 61.59 (10.979) | 55.68 (18.837)
  CD45+CD3-CD16+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 62.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.71 (10.282) | 52.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.29 (11.006) | 63.25 (9.771) | 58.44 (14.956)
  CD45+CD3-CD16+CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 65.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 57.62 (13.987) |  | 57.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD69+CD107-; D8; n=1,3,0,5,4,8 | 44.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.06 (8.555) |  | 58.99 (8.379) | 65.52 (2.097) | 43.74 (17.564)
  CD45+CD3-CD16+CD69+CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69+CD107-; D15;S1; n=1,3,1,5,4,9 | 64.68 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 71.45 (1.611) | 57.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.34 (4.338) | 63.57 (6.498) | 57.42 (15.273)
  CD45+CD3-CD16+CD69+CD107-; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+CD107-; D15; S2; n=0,0,1,0,0,0 |  |  | 27.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD69+CD107-; D29; n=1,3,1,4,4,8 | 62.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 73.22 (4.103) | 34.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.98 (6.511) | 55.64 (6.702) | 58.48 (19.691)
  CD45+CD3-CD16+CD69+CD107-; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD69+CD107-; FU; n=1,2,0,3,1,4 | 63.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.16 (15.047) |  | 50.46 (18.585) | 64.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 53.69 (9.671)
  CD45+CD3-CD16+CD69+CD107-; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69+CD107-; USC; n=0,0,1,0,0,0 |  |  | 49.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69-CD107+; D1;pre n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107+; D1;pre n=1,3,1,5,4,9 | 0.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.07 (0.115) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.22 (0.265) | 0.43 (0.395) | 0.36 (0.740)
  CD45+CD3-CD16+CD69-CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107+; D1;1 h;n=1,3,1,5,4,9 | 0.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.31 (0.399) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.14 (0.238) | 0.24 (0.441) | 0.32 (0.494)
  CD45+CD3-CD16+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.09 (0.162) | 2.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.05 (0.069) | 0.23 (0.403) | 0.48 (1.014)
  CD45+CD3-CD16+CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.54 (0.764) |  | 0.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD69-CD107+; D8; n=1,3,0,5,4,8 | 0.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.14 (0.029) |  | 0.07 (0.100) | 0.04 (0.041) | 0.66 (0.524)
  CD45+CD3-CD16+CD69-CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107+; D15;S1; n=1,3,1,5,4,9 | 0.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.12 (0.102) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.05 (0.121) | 0.19 (0.236) | 0.56 (0.890)
  CD45+CD3-CD16+CD69-CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69-CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 1.09 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD69-CD107+; D29; n=1,3,1,4,4,8 | 0.52 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.07 (0.127) | 2.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.32 (0.326) | 0.34 (0.241) | 1.14 (1.844)
  CD45+CD3-CD16+CD69-CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD69-CD107+; FU; n=1,2,0,3,1,4 | 0.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.26 (0.361) |  | 0.22 (0.333) | 0.09 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.27 (0.324)
  CD45+CD3-CD16+CD69-CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69-CD107+; USC; n=0,0,1,0,0,0 |  |  | 0.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69-CD107-; D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107-; D1;pre; n=1,3,1,5,4,9 | 31.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.57 (3.611) | 16.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.86 (7.256) | 17.07 (3.528) | 23.98 (15.442)
  CD45+CD3-CD16+CD69-CD107-; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107-; D1;1 h;n=1,3,1,5,4,9 | 22.68 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.93 (2.396) | 12.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.98 (8.736) | 13.75 (3.880) | 21.36 (16.671)
  CD45+CD3-CD16+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD16+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 22.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.91 (12.511) | 6.58 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.70 (5.783) | 15.21 (4.603) | 19.98 (11.842)
  CD45+CD3-CD16+CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD16+CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 9.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.43 (4.540) |  | 11.32 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD16+CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD16+CD69-CD107-; D8; n=1,3,0,5,4,8 | 21.78 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.03 (5.842) |  | 18.63 (10.331) | 20.05 (2.014) | 28.47 (21.443)
  CD45+CD3-CD16+CD69-CD107-; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD16+CD69-CD107-; D15; S1;n=1,3,1,5,4,9 | 18.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.84 (3.338) | 3.51 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.67 (6.810) | 18.13 (7.060) | 20.92 (19.349)
  CD45+CD3-CD16+CD69-CD107-; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69-CD107-; D15; S2; n=0,0,1,0,0,0 |  |  | 6.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD16+CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD16+CD69-CD107-; D29; n=1,3,1,4,4,8 | 20.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.00 (2.247) | 12.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.97 (6.747) | 16.67 (6.466) | 24.35 (16.239)
  CD45+CD3-CD16+CD69-CD107-; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD16+CD69-CD107-; FU; n=1,2,0,3,1,4 | 22.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.35 (1.146) |  | 18.34 (12.586) | 23.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.89 (19.247)
  CD45+CD3-CD16+CD69-CD107-; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD16+CD69-CD107-; USC; n=0,0,1,0,0,0 |  |  | 34.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+; D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+; D1;pre; n=1,3,1,5,4,9 | 67.22 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 78.33 (3.952) | 82.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.55 (7.943) | 77.94 (6.341) | 71.81 (14.980)
  CD45+CD3-CD56+CD69+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+; D1;1 h;n=1,3,1,5,4,9 | 75.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.13 (4.906) | 86.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.21 (8.936) | 80.38 (5.074) | 73.55 (18.249)
  CD45+CD3-CD56+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD69+;D1;6 h;n=1,3,1,5,4,11 | 79.56 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 74.82 (11.935) | 92.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.05 (5.668) | 79.33 (8.307) | 74.28 (14.068)
  CD45+CD3-CD56+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD69+; D2; n=0,0,1,2,0,1 |  |  | 87.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 84.69 (5.862) |  | 84.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD69+; D8; n=1,3,0,5,4,8 | 75.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.08 (3.948) |  | 77.49 (9.757) | 75.71 (6.039) | 64.20 (17.380)
  CD45+CD3-CD56+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+; D15;S1; n=1,3,1,5,4,9 | 80.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.83 (2.746) | 93.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.69 (5.772) | 77.05 (1.250) | 74.14 (18.976)
  CD45+CD3-CD56+CD69+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+; D15; S2; n=0,0,1,0,0,0 |  |  | 90.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD69+; D29; n=1,3,1,4,4,8 | 76.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.41 (3.445) | 83.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.90 (5.693) | 78.39 (3.376) | 72.21 (20.172)
  CD45+CD3-CD56+CD69+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD69+; FU; n=1,2,0,3,1,4 | 75.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 83.15 (0.643) |  | 78.85 (8.804) | 76.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 75.78 (15.172)
  CD45+CD3-CD56+CD69+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+; USC; n=0,0,1,0,0,0 |  |  | 64.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD107+; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD107+; D1; pre; n=1,3,1,5,4,9 | 2.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.70 (5.812) | 15.32 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.30 (12.987) | 20.36 (10.285) | 15.35 (12.755)
  CD45+CD3-CD56+CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD107+; D1;1 h;n=1,3,1,5,4,9 | 5.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.87 (7.853) | 6.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.11 (11.990) | 18.36 (8.295) | 13.92 (14.620)
  CD45+CD3-CD56+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD107+;D1;6 h;n=1,3,1,5,4,11 | 14.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.66 (7.368) | 31.76 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.41 (13.644) | 19.50 (10.930) | 17.82 (13.218)
  CD45+CD3-CD56+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD107+; D2; n=0,0,1,2,0,1 |  |  | 21.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 28.04 (7.347) |  | 26.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD107+; D8; n=1,3,0,5,4,8 | 32.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.79 (2.953) |  | 17.46 (7.730) | 12.81 (2.027) | 15.17 (12.783)
  CD45+CD3-CD56+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD107+; D15;S1; n=1,3,1,5,4,9 | 15.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.48 (3.558) | 39.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.18 (7.919) | 13.95 (4.221) | 16.02 (10.352)
  CD45+CD3-CD56+CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 54.4 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD107+; D29; n=1,3,1,4,4,8 | 15.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.77 (3.841) | 48.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.09 (1.735) | 22.89 (7.527) | 17.13 (5.406)
  CD45+CD3-CD56+CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD107+; FU; n=1,2,0,3,1,4 | 13.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.93 (11.469) |  | 26.54 (22.053) | 11.46 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.63 (17.232)
  CD45+CD3-CD56+CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD107+; USC; n=0,0,1,0,0,0 |  |  | 16.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+CD107+; D1; pre n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107+; D1; pre n=1,3,1,5,4,9 | 2.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.58 (5.907) | 15.32 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.98 (12.746) | 19.90 (9.878) | 15.06 (12.804)
  CD45+CD3-CD56+CD69+CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107+; D1;1 h;n=1,3,1,5,4,9 | 4.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.56 (7.455) | 6.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.90 (11.974) | 17.72 (8.423) | 13.60 (14.641)
  CD45+CD3-CD56+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 14.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.94 (6.586) | 31.76 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.27 (13.781) | 19.15 (10.796) | 15.67 (9.351)
  CD45+CD3-CD56+CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 21.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.36 (7.460) |  | 25.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD69+CD107+; D8; n=1,3,0,5,4,8 | 31.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.63 (2.770) |  | 17.32 (7.645) | 12.69 (2.047) | 14.33 (12.481)
  CD45+CD3-CD56+CD69+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107+; D15;S1; n=1,3,1,5,4,9 | 15.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.40 (3.545) | 39.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.03 (7.922) | 13.80 (4.123) | 15.58 (10.540)
  CD45+CD3-CD56+CD69+CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 54.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD69+CD107+; D29; n=1,3,1,4,4,8 | 15.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.77 (3.841) | 46.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.70 (1.922) | 22.55 (7.441) | 15.59 (4.963)
  CD45+CD3-CD56+CD69+CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD69+CD107+; FU; n=1,2,0,3,1,4 | 13.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.60 (11.130) |  | 26.27 (22.189) | 11.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.00 (16.629)
  CD45+CD3-CD56+CD69+CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+CD107+; USC; n=0,0,1,0,0,0 |  |  | 15.52 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+CD107-; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107-; D1; pre; n=1,3,1,5,4,9 | 64.78 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 66.74 (7.360) | 66.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.56 (9.286) | 58.04 (12.938) | 56.75 (10.180)
  CD45+CD3-CD56+CD69+CD107-; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107-; D1;1 h;n=1,3,1,5,4,9 | 70.36 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.58 (7.453) | 80.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.31 (7.582) | 62.66 (8.744) | 59.95 (15.044)
  CD45+CD3-CD56+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 64.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 58.88 (10.865) | 61.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 56.78 (8.650) | 60.18 (9.203) | 58.62 (14.204)
  CD45+CD3-CD56+CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 65.83 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 57.33 (13.329) |  | 58.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD69+CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69+CD107-; D15;S1; n=1,3,1,5,4,9 | 64.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.43 (0.830) | 54.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.66 (4.313) | 63.25 (5.044) | 58.55 (14.595)
  CD45+CD3-CD56+CD69+CD107-; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+CD107-; D15; S2; n=0,0,1,0,0,0 |  |  | 36.52 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD69+CD107-; D8; n=1,3,0,5,4,8 | 44.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.44 (6.176) |  | 60.18 (8.140) | 63.02 (5.005) | 49.87 (13.422)
  CD45+CD3-CD56+CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD69+CD107-; D29; n=1,3,1,4,4,8 | 61.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.64 (2.420) | 36.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.21 (4.900) | 55.84 (6.851) | 56.62 (21.533)
  CD45+CD3-CD56+CD69+CD107-; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD69+CD107-; FU; n=1,2,0,3,1,4 | 62.71 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.55 (11.780) |  | 52.58 (16.165) | 65.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.78 (12.864)
  CD45+CD3-CD56+CD69+CD107-; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69+CD107-; USC; n=0,0,1,0,0,0 |  |  | 49.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69-CD107+; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107+; D1; pre; n=1,3,1,5,4,9 | 0.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.11 (0.095) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.31 (0.267) | 0.46 (0.425) | 0.29 (0.558)
  CD45+CD3-CD56+CD69-CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107+; D1;1 h;n=1,3,1,5,4,9 | 0.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.31 (0.412) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.21 (0.123) | 0.64 (0.660) | 0.32 (0.364)
  CD45+CD3-CD56+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.72 (0.968) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.14 (0.226) | 0.35 (0.262) | 2.15 (5.749)
  CD45+CD3-CD56+CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.68 (0.113) |  | 0.46 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD69-CD107+; D8; n=1,3,0,5,4,8 | 1.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.16 (0.182) |  | 0.14 (0.186) | 0.11 (0.109) | 0.84 (1.031)
  CD45+CD3-CD56+CD69-CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107+; D15;S1; n=1,3,1,5,4,9 | 0.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.09 (0.076) | 0 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.15 (0.145) | 0.15 (0.174) | 0.44 (0.638)
  CD45+CD3-CD56+CD69-CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69-CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 0.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD69-CD107+; D29; n=1,3,1,4,4,8 | 0.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.00 (0.000) | 1.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.39 (0.541) | 0.35 (0.145) | 1.54 (2.079)
  CD45+CD3-CD56+CD69-CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD69-CD107+; FU; n=1,2,0,3,1,4 | 0.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.34 (0.332) |  | 0.27 (0.379) | 0.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.62 (0.678)
  CD45+CD3-CD56+CD69-CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69-CD107+; USC; n=0,0,1,0,0,0 |  |  | 0.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69-CD107-; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107-; D1; pre; n=1,3,1,5,4,9 | 32.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.56 (3.938) | 17.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.14 (8.116) | 21.60 (6.379) | 27.91 (14.759)
  CD45+CD3-CD56+CD69-CD107-; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107-; D1;1 h;n=1,3,1,5,4,9 | 24.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.55 (5.154) | 13.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.58 (8.921) | 18.99 (4.842) | 26.13 (18.140)
  CD45+CD3-CD56+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 20.44 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.46 (11.748) | 7.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.81 (5.486) | 20.36 (8.302) | 23.56 (13.128)
  CD45+CD3-CD56+CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 12.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.64 (5.975) |  | 14.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD69-CD107-; D8; n=1,3,0,5,4,8 | 23.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.76 (3.835) |  | 22.37 (9.797) | 24.18 (5.949) | 34.96 (16.868)
  CD45+CD3-CD56+CD69-CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD69-CD107-; D15;S1; n=1,3,1,5,4,9 | 19.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.09 (2.774) | 6.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.16 (5.735) | 22.81 (1.095) | 25.43 (18.427)
  CD45+CD3-CD56+CD69-CD107-; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69-CD107-; D15; S2; n=0,0,1,0,0,0 |  |  | 9.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD69-CD107-; D29; n=1,3,1,4,4,8 | 22.56 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.59 (3.445) | 14.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.73 (5.751) | 21.27 (3.470) | 26.26 (18.208)
  CD45+CD3-CD56+CD69-CD107-; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD69-CD107-; FU; n=1,2,0,3,1,4 | 24.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.52 (0.311) |  | 20.87 (8.475) | 23.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.60 (15.370)
  CD45+CD3-CD56+CD69-CD107-; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD69-CD107-; USC; n=0,0,1,0,0,0 |  |  | 34.48 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD16+CD69+; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD69+; D1; pre; n=1,3,1,5,4,9 | 67.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.63 (3.253) | 83.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.66 (7.578) | 82.35 (3.605) | 75.53 (16.495)
  CD45+CD3-CD56+CD16+CD69+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD69+; D1;1 h;n=1,3,1,5,4,9 | 76.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.33 (2.688) | 88.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 81.64 (9.116) | 85.57 (3.640) | 77.45 (18.036)
  CD45+CD3-CD56+CD16+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD16+CD69+;D1;6 h;n=1,3,1,5,4,11 | 78.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.67 (11.942) | 93.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 83.35 (5.763) | 83.95 (4.687) | 78.92 (13.044)
  CD45+CD3-CD56+CD16+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD16+CD69+; D2; n=0,0,1,2,0,1 |  |  | 90.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 89.13 (3.147) |  | 87.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD16+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD16+CD69+; D8; n=1,3,0,5,4,8 | 77.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 75.37 (5.656) |  | 80.55 (10.272) | 79.75 (2.003) | 70.62 (21.607)
  CD45+CD3-CD56+CD16+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD69+; D15;S1; n=1,3,1,5,4,9 | 81.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 78.47 (3.127) | 97.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.94 (6.952) | 80.67 (5.845) | 79.09 (19.651)
  CD45+CD3-CD56+CD16+CD69+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD16+CD69+; D15; S2; n=0,0,1,0,0,0 |  |  | 94.42 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD16+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD16+CD69+; D29; n=1,3,1,4,4,8 | 78.98 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 81.90 (2.566) | 85.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.16 (7.448) | 82.36 (4.976) | 74.62 (18.799)
  CD45+CD3-CD56+CD16+CD69+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD16+CD69+; FU; n=1,2,0,3,1,4 | 77.43 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 83.80 (1.485) |  | 81.09 (12.356) | 76.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 80.93 (19.159)
  CD45+CD3-CD56+CD16+CD69+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD16+CD69+; USC; n=0,0,1,0,0,0 |  |  | 65.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD16+CD107+; D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD107+; D1;pre; n=1,3,1,5,4,9 | 6.82 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.17 (5.660) | 16.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.55 (13.586) | 22.71 (12.190) | 23.18 (31.567)
  CD45+CD3-CD56+CD16+CD107+; D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD107+; D1;1 h;n=1,3,1,5,4,9 | 12.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.37 (7.788) | 7.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.24 (13.929) | 23.33 (14.182) | 20.40 (26.478)
  CD45+CD3-CD56+CD16+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD56+CD16+CD107+;D1;6 h;n=1,3,1,5,4,11 | 15.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.86 (7.082) | 31.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.52 (16.167) | 20.47 (12.384) | 19.35 (17.934)
  CD45+CD3-CD56+CD16+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD56+CD16+CD107+; D2; n=0,0,1,2,0,1 |  |  | 25.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 32.24 (9.970) |  | 30.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD56+CD16+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD56+CD16+CD107+; D8; n=1,3,0,5,4,8 | 33.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.53 (3.339) |  | 18.59 (9.084) | 13.90 (2.089) | 26.69 (33.377)
  CD45+CD3-CD56+CD16+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD56+CD16+CD107+; D15;S1; n=1,3,1,5,4,9 | 16.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.20 (4.025) | 40.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.69 (8.825) | 14.72 (4.613) | 21.04 (17.138)
  CD45+CD3-CD56+CD16+CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD16+CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 60.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD56+CD16+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD56+CD16+CD107+; D29; n=1,3,1,4,4,8 | 16.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.01 (4.316) | 50.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.68 (2.613) | 25.75 (9.873) | 18.09 (7.210)
  CD45+CD3-CD56+CD16+CD107+; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD56+CD16+CD107+; FU; n=1,2,0,3,1,4 | 13.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.58 (14.078) |  | 29.76 (28.400) | 11.68 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.61 (14.702)
  CD45+CD3-CD56+CD16+CD107+; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD56+CD16+CD107+; USC; n=0,0,1,0,0,0 |  |  | 16.42 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX241; D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX241; D1;pre; n=1,3,1,5,4,9 | 6.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.09 (5.664) | 16.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.32 (13.319) | 22.27 (11.808) | 22.97 (31.676)
  CDX241; D1;1h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX241; D1;1h;n=1,3,1,5,4,9 | 12.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.02 (7.382) | 7.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.15 (13.818) | 23.12 (14.060) | 20.23 (26.492)
  CDX241; D1;6h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CDX241; D1;6h;n=1,3,1,5,4,11 | 15.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.75 (6.934) | 31.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.46 (16.219) | 20.23 (12.033) | 19.06 (18.044)
  CDX241; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CDX241; D2; n=0,0,1,2,0,1 |  |  | 25.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.68 (10.769) |  | 29.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CDX241; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CDX241; D8; n=1,3,0,5,4,8 | 32.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.47 (3.238) |  | 18.50 (9.029) | 13.88 (2.075) | 26.20 (33.362)
  CDX241; D15;S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX241; D15;S1;n=1,3,1,5,4,9 | 15.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.13 (3.908) | 40.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.62 (8.827) | 14.55 (4.521) | 20.62 (17.353)
  CDX241; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX241; D15;S2; n=0,0,1,0,0,0 |  |  | 60.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX241; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CDX241; D29; n=1,3,1,4,4,8 | 15.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.01 (4.316) | 49.39 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.40 (2.640) | 25.56 (9.917) | 16.64 (6.597)
  CDX241; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CDX241; FU; n=1,2,0,3,1,4 | 13.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.29 (13.668) |  | 29.58 (28.512) | 11.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.41 (14.820)
  CDX241; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX241; USC; n=0,0,1,0,0,0 |  |  | 15.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX243; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX243; D1; pre; n=1,3,1,5,4,9 | 61.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.54 (8.092) | 66.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.34 (9.199) | 60.08 (11.697) | 52.56 (22.645)
  CDX243; D1;1h; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX243; D1;1h; n=1,3,1,5,4,9 | 64.84 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.31 (7.929) | 80.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.49 (8.086) | 62.45 (11.395) | 57.22 (19.058)
  CDX243;D1;6h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CDX243;D1;6h; n=1,3,1,5,4,11 | 63.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.93 (9.710) | 61.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.89 (11.139) | 63.72 (9.993) | 59.86 (14.378)
  CDX243; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CDX243; D2; n=0,0,1,2,0,1 |  |  | 65.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 57.46 (13.909) |  | 57.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CDX243; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CDX243; D8; n=1,3,0,5,4,8 | 44.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.91 (8.623) |  | 62.04 (7.093) | 65.87 (2.821) | 44.43 (22.911)
  CDX243; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX243; D15;S1; n=1,3,1,5,4,9 | 65.55 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.34 (0.958) | 56.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.32 (4.554) | 66.13 (9.524) | 58.47 (16.070)
  CDX243; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX243; D15;S2; n=0,0,1,0,0,0 |  |  | 33.48 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX243; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CDX243; D29; n=1,3,1,4,4,8 | 62.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 73.88 (3.073) | 36.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.75 (5.261) | 56.80 (5.697) | 57.98 (21.467)
  CDX243; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CDX243; FU;n=1,2,0,3,1,4 | 63.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.51 (15.146) |  | 51.52 (18.071) | 65.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.52 (9.421)
  CDX243; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX243; USC;n=0,0,1,0,0,0 |  |  | 49.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX244; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX244; D1; pre; n=1,3,1,5,4,9 | 0.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.08 (0.139) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.23 (0.289) | 0.45 (0.422) | 0.21 (0.505)
  CDX244; D1;1h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX244; D1;1h;n=1,3,1,5,4,9 | 0.39 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.35 (0.454) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.09 (0.137) | 0.22 (0.391) | 0.17 (0.319)
  CDX244; D1;6h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CDX244; D1;6h;n=1,3,1,5,4,11 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.11 (0.191) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.06 (0.089) | 0.24 (0.423) | 0.30 (0.682)
  CDX244; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CDX244; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.57 (0.799) |  | 0.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CDX244; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CDX244; D8; n=1,3,0,5,4,8 | 0.98 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.06 (0.110) |  | 0.08 (0.116) | 0.02 (0.045) | 0.49 (0.601)
  CDX244; D15;S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX244; D15;S1;n=1,3,1,5,4,9 | 0.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.07 (0.115) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.71 (0.204) | 0.42 (0.632)
  CDX244; D15;S2n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX244; D15;S2n=0,0,1,0,0,0 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX244; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CDX244; D29; n=1,3,1,4,4,8 | 0.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.00 (0.000) | 1.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.28 (0.392) | 0.19 (0.194) | 1.46 (1.849)
  CDX244; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CDX244; FU;n=1,2,0,3,1,4 | 0.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.29 (0.410) |  | 0.18 (0.267) | 0.09 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.20 (0.189)
  CDX244; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX244; USC;n=0,0,1,0,0,0 |  |  | 0.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX245; D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX245; D1; pre; n=1,3,1,5,4,9 | 31.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.28 (3.144) | 16.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.11 (7.819) | 17.21 (3.797) | 24.26 (16.218)
  CDX245; D1; 1h; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX245; D1; 1h; n=1,3,1,5,4,9 | 22.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.32 (2.902) | 11.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.27 (9.233) | 14.21 (3.682) | 22.37 (17.894)
  CDX245; D1; 6h; n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CDX245; D1; 6h; n=1,3,1,5,4,11 | 21.76 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.22 (11.931) | 6.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.59 (5.742) | 15.82 (4.876) | 20.79 (12.726)
  CDX245; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CDX245; D2; n=0,0,1,2,0,1 |  |  | 9.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.31 (3.946) |  | 11.46 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CDX245; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CDX245; D8; n=1,3,0,5,4,8 | 22.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.56 (5.547) |  | 19.37 (10.290) | 20.23 (1.977) | 28.88 (21.510)
  CDX245; D15; S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CDX245; D15; S1; n=1,3,1,5,4,9 | 18.22 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.46 (3.242) | 2.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.00 (6.887) | 19.16 (5.695) | 20.48 (19.116)
  CDX245; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX245; D15; S2; n=0,0,1,0,0,0 |  |  | 5.58 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CDX245; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CDX245; D29; n=1,3,1,4,4,8 | 20.48 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.10 (2.566) | 12.58 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.57 (7.550) | 17.45 (4.991) | 23.93 (16.995)
  CDX245; FU; n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CDX245; FU; n=1,2,0,3,1,4 | 22.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.91 (1.075) |  | 18.72 (12.153) | 23.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.88 (18.996)
  CDX245; USC; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CDX245; USC; n=0,0,1,0,0,0 |  |  | 33.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+;D1pre; n=1,3,1,5,4,9 | 62.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.83 (5.748) | 84.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.05 (13.328) | 80.50 (5.553) | 72.52 (20.777)
  CD45+CD3+CD56+CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+;D1;1 h;n=1,3,1,5,4,9 | 71.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.91 (8.757) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 74.68 (12.530) | 76.76 (7.819) | 69.96 (23.711)
  CD45+CD3+CD56+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD69+;D1;6 h;n=1,3,1,5,4,11 | 77.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.55 (11.000) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 75.64 (10.831) | 77.96 (9.405) | 73.92 (20.707)
  CD45+CD3+CD56+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD69+; D2; n=0,0,1,2,0,1 |  |  | 90.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.51 (11.823) |  | 81.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD69+; D8; n=1,3,0,5,4,8 | 70.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 79.41 (6.359) |  | 77.26 (8.083) | 77.76 (3.671) | 71.42 (17.583)
  CD45+CD3+CD56+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+; D15;S1; n=1,3,1,5,4,9 | 76.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 81.26 (7.195) | 100 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 76.72 (9.716) | 75.78 (3.311) | 72.29 (22.078)
  CD45+CD3+CD56+CD69+;D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+;D15;S2; n=0,0,1,0,0,0 |  |  | 90.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD69+; D29; n=1,3,1,4,4,8 | 76.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 84.46 (9.848) | 92.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 75.11 (5.695) | 79.47 (4.516) | 73.25 (19.837)
  CD45+CD3+CD56+CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD69+; FU;n=1,2,0,3,1,4 | 76.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 83.76 (2.977) |  | 76.93 (2.841) | 78.84 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 78.73 (13.208)
  CD45+CD3+CD56+CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+; USC;n=0,0,1,0,0,0 |  |  | 73.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD107+;D1pre; n=1,3,1,5,4,9 | 8.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.44 (3.025) | 30.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.69 (14.219) | 25.59 (10.582) | 21.94 (11.569)
  CD45+CD3+CD56+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD107+;D1;1 h;n=1,3,1,5,4,9 | 16.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.59 (8.435) | 16.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.84 (13.782) | 20.17 (7.408) | 19.38 (9.838)
  CD45+CD3+CD56+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD107+;D1;6 h;n=1,3,1,5,4,11 | 17.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.55 (9.084) | 77.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.54 (14.785) | 18.38 (7.558) | 27.83 (16.580)
  CD45+CD3+CD56+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD107+; D2; n=0,0,1,2,0,1 |  |  | 50.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.40 (2.892) |  | 21.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD107+; D8; n=1,3,0,5,4,8 | 34.51 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.08 (12.140) |  | 22.70 (6.042) | 23.85 (15.031) | 25.37 (9.055)
  CD45+CD3+CD56+CD107+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD107+; D15; S1;n=1,3,1,5,4,9 | 24.44 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.39 (9.804) | 66.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.15 (15.543) | 22.75 (9.361) | 24.77 (13.389)
  CD45+CD3+CD56+CD107+;D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD107+;D15;S2; n=0,0,1,0,0,0 |  |  | 91.36 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD107+; D29; n=1,3,1,4,4,8 | 19.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.61 (12.809) | 94.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.97 (16.720) | 26.64 (16.501) | 25.47 (7.825)
  CD45+CD3+CD56+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD107+; FU;n=1,2,0,3,1,4 | 19.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.79 (8.132) |  | 32.87 (23.340) | 16.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 26.92 (16.312)
  CD45+CD3+CD56+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD107+; USC;n=0,0,1,0,0,0 |  |  | 20.51 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+CD107+;D1;pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107+;D1;pre; n=1,3,1,5,4,9 | 8.10 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.26 (2.974) | 30.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.85 (14.628) | 24.97 (10.148) | 21.16 (11.995)
  CD45+CD3+CD56+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9 | 15.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 25.29 (8.566) | 16.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.96 (14.211) | 19.58 (6.559) | 18.93 (9.947)
  CD45+CD3+CD56+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 17.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 26.84 (8.938) | 77.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.77 (15.022) | 17.89 (7.034) | 26.49 (16.563)
  CD45+CD3+CD56+CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 50.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.24 (3.111) |  | 20.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD69+CD107+; D8; n=1,3,0,5,4,8 | 32.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.24 (11.427) |  | 22.33 (5.946) | 23.10 (14.534) | 24.68 (9.353)
  CD45+CD3+CD56+CD69+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107+; D15;S1; n=1,3,1,5,4,9 | 24.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.22 (9.646) | 66.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.78 (15.294) | 22.25 (9.194) | 23.91 (13.531)
  CD45+CD3+CD56+CD69+CD107+;D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+CD107+;D15;S2; n=0,0,1,0,0,0 |  |  | 85.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD69+CD107+; D29; n=1,3,1,4,4,8 | 18.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.31 (12.597) | 86.84 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.41 (16.520) | 25.87 (15.887) | 23.72 (7.717)
  CD45+CD3+CD56+CD69+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD69+CD107+; FU;n=1,2,0,3,1,4 | 19.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.48 (8.217) |  | 31.89 (22.622) | 15.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 26.51 (16.034)
  CD45+CD3+CD56+CD69+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+CD107+; USC;n=0,0,1,0,0,0 |  |  | 16.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+CD107-;D1; pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107-;D1; pre; n=1,3,1,5,4,9 | 54.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 54.57 (2.810) | 53.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.20 (11.519) | 55.53 (15.219) | 51.35 (15.196)
  CD45+CD3+CD56+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9 | 56.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.62 (3.308) | 83.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 49.72 (10.923) | 57.19 (10.200) | 51.04 (17.281)
  CD45+CD3+CD56+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 60.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 49.71 (2.501) | 22.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.88 (11.326) | 60.07 (13.763) | 47.43 (15.287)
  CD45+CD3+CD56+CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 40.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.28 (8.719) |  | 60.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD69+CD107-; D8; n=1,3,0,5,4,8 | 38.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.17 (6.740) |  | 54.92 (10.367) | 54.67 (12.323) | 46.74 (9.237)
  CD45+CD3+CD56+CD69+CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69+CD107-; D15;S1; n=1,3,1,5,4,9 | 52.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.04 (6.660) | 33.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 56.94 (9.081) | 53.53 (10.408) | 48.38 (17.947)
  CD45+CD3+CD56+CD69+CD107-;D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+CD107-;D15;S2;n=0,0,1,0,0,0 |  |  | 5.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD69+CD107-; D29; n=1,3,1,4,4,8 | 57.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.14 (4.928) | 5.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 53.70 (12.139) | 53.61 (15.433) | 49.53 (16.556)
  CD45+CD3+CD56+CD69+CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD69+CD107-; FU;n=1,2,0,3,1,4 | 57.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 56.28 (5.240) |  | 45.05 (22.028) | 62.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.22 (5.130)
  CD45+CD3+CD56+CD69+CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69+CD107-; USC;n=0,0,1,0,0,0 |  |  | 56.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69-CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107+;D1pre; n=1,3,1,5,4,9 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.19 (0.163) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.84 (1.119) | 0.62 (0.761) | 0.77 (1.157)
  CD45+CD3+CD56+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9 | 1.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.30 (0.295) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.87 (1.493) | 0.59 (0.889) | 0.45 (0.501)
  CD45+CD3+CD56+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.72 (0.806) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.77 (1.369) | 0.49 (0.666) | 1.35 (2.225)
  CD45+CD3+CD56+CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.16 (0.219) |  | 0.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD69-CD107+; D8; n=1,3,0,5,4,8 | 2.43 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.84 (0.716) |  | 0.37 (0.613) | 0.75 (0.573) | 0.69 (0.656)
  CD45+CD3+CD56+CD69-CD107+; D15;S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107+; D15;S1;n=1,3,1,5,4,9 | 0.32 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.17 (0.300) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.37 (0.288) | 0.51 (0.307) | 0.87 (1.194)
  CD45+CD3+CD56+CD69-CD107+;D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69-CD107+;D15;S2;n=0,0,1,0,0,0 |  |  | 5.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD69-CD107+; D29; n=1,3,1,4,4,8 | 0.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.29 (0.409) | 7.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.57 (0.312) | 0.77 (0.697) | 1.75 (2.925)
  CD45+CD3+CD56+CD69-CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD69-CD107+; FU;n=1,2,0,3,1,4 | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.31 (0.085) |  | 0.98 (1.235) | 0.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.41 (0.407)
  CD45+CD3+CD56+CD69-CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69-CD107+; USC;n=0,0,1,0,0,0 |  |  | 3.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69-CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107-;D1pre; n=1,3,1,5,4,9 | 37.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.98 (5.814) | 15.38 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.11 (12.486) | 18.88 (5.007) | 26.71 (19.740)
  CD45+CD3+CD56+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9 | 27.78 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.78 (8.736) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.444 (11.410) | 22.65 (7.631) | 29.59 (23.473)
  CD45+CD3+CD56+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD56+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 22.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.74 (11.250) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.59 (9.836) | 21.55 (8.954) | 24.74 (19.457)
  CD45+CD3+CD56+CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD56+CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 10.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.34 (11.604) |  | 18.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD56+CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD56+CD69-CD107-; D8; n=1,3,0,5,4,8 | 27.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.75 (7.018) |  | 22.38 (7.709) | 21.49 (4.140) | 27.89 (17.180)
  CD45+CD3+CD56+CD69-CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD56+CD69-CD107-; D15;S1; n=1,3,1,5,4,9 | 23.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.56 (7.134) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.91 (9.852) | 23.72 (3.040) | 26.84 (21.388)
  CD45+CD3+CD56+CD69-CD107-;D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69-CD107-;D15;S2;n=0,0,1,0,0,0 |  |  | 3.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD56+CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD56+CD69-CD107-; D29; n=1,3,1,4,4,8 | 22.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.25 (9.918) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.33 (5.914) | 19.76 (4.920) | 25.00 (18.022)
  CD45+CD3+CD56+CD69-CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD56+CD69-CD107-; FU;n=1,2,0,3,1,4 | 23.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 15.94 (2.892) |  | 22.09 (2.249) | 20.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.86 (13.394)
  CD45+CD3+CD56+CD69-CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD56+CD69-CD107-; USC;n=0,0,1,0,0,0 |  |  | 23.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+;D1pre; n=1,3,1,5,4,9 | 57.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 71.12 (1.083) | 59.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.19 (9.089) | 69.48 (7.473) | 64.41 (15.841)
  CD45+CD3+CD8+CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+;D1;1 h;n=1,3,1,5,4,9 | 54.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 66.55 (0.781) | 66.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.39 (8.060) | 69.27 (10.664) | 62.62 (18.568)
  CD45+CD3+CD8+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD69+;D1;6 h;n=1,3,1,5,4,11 | 70.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.77 (2.867) | 81.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.66 (7.411) | 69.44 (10.476) | 64.10 (16.568)
  CD45+CD3+CD8+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD69+; D2; n=0,0,1,2,0,1 |  |  | 71.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 77.60 (7.898) |  | 73.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD69+; D8; n=1,3,0,5,4,8 | 63.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.38 (2.682) |  | 71.51 (5.945) | 69.15 (2.032) | 59.81 (14.230)
  CD45+CD3+CD8+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+; D15;S1; n=1,3,1,5,4,9 | 66.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.12 (3.641) | 67.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.11 (5.807) | 65.46 (2.301) | 58.44 (20.646)
  CD45+CD3+CD8+CD69+; D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+; D15;S2;n=0,0,1,0,0,0 |  |  | 69.60 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD69+; D29; n=1,3,1,4,4,8 | 68.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.13 (0.599) | 52.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.07 (4.666) | 70.42 (3.658) | 60.96 (16.314)
  CD45+CD3+CD8+CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD69+; FU;n=1,2,0,3,1,4 | 67.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 74.76 (3.903) |  | 74.36 (3.927) | 70.80 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.63 (13.052)
  CD45+CD3+CD8+CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+; USC;n=0,0,1,0,0,0 |  |  | 45.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD107+;D1pre; n=1,3,1,5,4,9 | 9.25 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.58 (6.553) | 17.31 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.38 (10.840) | 19.50 (5.678) | 12.96 (7.622)
  CD45+CD3+CD8+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD107+;D1;1 h;n=1,3,1,5,4,9 | 11.02 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.64 (7.885) | 4.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.87 (10.264) | 17.86 (7.915) | 12.10 (9.816)
  CD45+CD3+CD8+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD107+;D1;6 h;n=1,3,1,5,4,11 | 13.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.21 (5.668) | 35.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.61 (12.241) | 17.74 (6.679) | 14.58 (7.973)
  CD45+CD3+CD8+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD107+; D2; n=0,0,1,2,0,1 |  |  | 25.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.03 (4.907) |  | 15.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD107+; D8; n=1,3,0,5,4,8 | 37.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 19.18 (3.660) |  | 24.12 (11.200) | 19.58 (10.034) | 13.53 (7.177)
  CD45+CD3+CD8+CD107+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD107+; D15; S1;n=1,3,1,5,4,9 | 20.58 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.59 (2.973) | 93.55 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 21.11 (14.964) | 18.52 (6.515) | 14.52 (11.560)
  CD45+CD3+CD8+CD107+; D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD107+; D15;S2;n=0,0,1,0,0,0 |  |  | 90.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD107+; D29; n=1,3,1,4,4,8 | 44.48 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.53 (2.105) | 66.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.44 (12.685) | 22.28 (10.800) | 16.01 (7.377)
  CD45+CD3+CD8+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD107+; FU;n=1,2,0,3,1,4 | 21.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.00 (7.545) |  | 34.50 (27.190) | 20.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.54 (20.530)
  CD45+CD3+CD8+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD107+; USC;n=0,0,1,0,0,0 |  |  | 13.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107+;D1pre; n=1,3,1,5,4,9 | 8.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.82 (6.136) | 16.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.35 (10.595) | 18.89 (5.513) | 12.42 (7.519)
  CD45+CD3+CD8+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9 | 10.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.60 (7.232) | 4.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 23.63 (10.069) | 17.10 (7.592) | 11.51 (9.671)
  CD45+CD3+CD8+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 13.70 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.92 (4.681) | 35.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.61 (11.463) | 16.83 (6.502) | 13.49 (8.242)
  CD45+CD3+CD8+CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 25.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.67 (4.391) |  | 15.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD69+CD107+; D8; n=1,3,0,5,4,8 | 33.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.86 (1.989) |  | 23.15 (10.176) | 18.62 (9.229) | 12.58 (6.811)
  CD45+CD3+CD8+CD69+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107+; D15;S1; n=1,3,1,5,4,9 | 19.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.35 (2.815) | 64.52 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.62 (14.511) | 17.46 (5.818) | 13.79 (11.461)
  CD45+CD3+CD8+CD69+CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 66.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD69+CD107+; D29; n=1,3,1,4,4,8 | 36.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 18.16 (2.172) | 44.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 17.79 (12.221) | 21.18 (9.942) | 14.79 (7.086)
  CD45+CD3+CD8+CD69+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD69+CD107+; FU;n=1,2,0,3,1,4 | 20.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.43 (7.177) |  | 33.05 (25.896) | 20.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.91 (18.370)
  CD45+CD3+CD8+CD69+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+CD107+; USC;n=0,0,1,0,0,0 |  |  | 12.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107-;D1pre; n=1,3,1,5,4,9 | 48.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 47.30 (5.590) | 43.27 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 46.85 (9.558) | 50.59 (11.155) | 51.99 (13.129)
  CD45+CD3+CD8+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9 | 44.32 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 45.95 (6.784) | 62.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 44.76 (7.470) | 52.17 (7.570) | 51.12 (15.653)
  CD45+CD3+CD8+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 56.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 43.85 (7.548) | 45.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 47.05 (7.908) | 52.61 (7.942) | 50.61 (11.996)
  CD45+CD3+CD8+CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 46.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.93 (12.282) |  | 57.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD69+CD107-; D8; n=1,3,0,5,4,8 | 29.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 47.53 (4.483) |  | 48.36 (11.067) | 50.52 (8.995) | 47.22 (12.334)
  CD45+CD3+CD8+CD69+CD107-; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69+CD107-; D15; S1;n=1,3,1,5,4,9 | 46.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 58.77 (6.439) | 3.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 51.49 (9.965) | 47.99 (7.314) | 44.65 (18.062)
  CD45+CD3+CD8+CD69+CD107-; D15; S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+CD107-; D15; S2;n=0,0,1,0,0,0 |  |  | 2.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD69+CD107-; D29; n=1,3,1,4,4,8 | 31.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 53.96 (1.639) | 7.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.28 (9.182) | 49.25 (12.319) | 46.17 (14.907)
  CD45+CD3+CD8+CD69+CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD69+CD107-; FU;n=1,2,0,3,1,4 | 47.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.34 (3.274) |  | 41.31 (23.301) | 50.44 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 47.72 (13.474)
  CD45+CD3+CD8+CD69+CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69+CD107-; USC;n=0,0,1,0,0,0 |  |  | 32.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69-CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107+;D1pre; n=1,3,1,5,4,9 | 0.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.76 (0.475) | 0.96 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.03 (1.228) | 0.61 (0.493) | 0.54 (0.575)
  CD45+CD3+CD8+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9 | 0.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.03 (0.683) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.24 (1.342) | 0.76 (0.919) | 0.59 (0.605)
  CD45+CD3+CD8+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.30 (1.040) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.01 (1.572) | 0.91 (0.629) | 1.09 (1.070)
  CD45+CD3+CD8+CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD69-CD107+; D8; n=1,3,0,5,4,8 | 4.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.32 (1.711) |  | 0.97 (1.172) | 0.96 (1.007) | 0.95 (1.058)
  CD45+CD3+CD8+CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.37 (0.516) |  | 0.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD69-CD107+; D15;S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107+; D15;S1;n=1,3,1,5,4,9 | 1.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.24 (0.163) | 29.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.48 (0.609) | 1.05 (0.920) | 0.73 (0.435)
  CD45+CD3+CD8+CD69-CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69-CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 23.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD69-CD107+; D29; n=1,3,1,4,4,8 | 7.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.37 (0.078) | 21.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.65 (0.554) | 1.10 (0.919) | 1.22 (1.347)
  CD45+CD3+CD8+CD69-CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD69-CD107+; FU;n=1,2,0,3,1,4 | 0.82 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.58 (0.361) |  | 1.44 (1.298) | 0.29 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.63 (2.326)
  CD45+CD3+CD8+CD69-CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69-CD107+; USC;n=0,0,1,0,0,0 |  |  | 1.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69-CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107-;D1pre; n=1,3,1,5,4,9 | 41.83 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 28.12 (1.219) | 39.42 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 28.78 (8.425) | 29.92 (7.082) | 35.04 (15.444)
  CD45+CD3+CD8+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9 | 44.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 32.42 (1.397) | 33.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 30.37 (7.516) | 29.97 (10.290) | 36.79 (18.243)
  CD45+CD3+CD8+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 29.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 33.94 (1.914) | 18.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.34 (7.255) | 29.65 (10.132) | 34.81 (15.738)
  CD45+CD3+CD8+CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8+CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 28.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.04 (7.382) |  | 26.77 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8+CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8+CD69-CD107-; D8; n=1,3,0,5,4,8 | 32.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 33.30 (2.044) |  | 27.52 (6.239) | 29.90 (2.006) | 39.24 (13.864)
  CD45+CD3+CD8+CD69-CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8+CD69-CD107-; D15;S1; n=1,3,1,5,4,9 | 32.56 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 29.64 (3.488) | 3.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.41 (6.016) | 33.49 (1.695) | 40.83 (20.434)
  CD45+CD3+CD8+CD69-CD107-; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69-CD107-; D15;S2; n=0,0,1,0,0,0 |  |  | 7.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8+CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8+CD69-CD107-; D29; n=1,3,1,4,4,8 | 23.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.50 (0.558) | 26.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.28 (4.954) | 28.48 (3.302) | 37.82 (15.640)
  CD45+CD3+CD8+CD69-CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8+CD69-CD107-; FU;n=1,2,0,3,1,4 | 31.20 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 24.67 (4.264) |  | 24.19 (5.014) | 28.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 27.74 (14.176)
  CD45+CD3+CD8+CD69-CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8+CD69-CD107-; USC;n=0,0,1,0,0,0 |  |  | 53.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+;D1pre; n=1,3,1,5,4,9 | 49.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.40 (2.410) | 61.84 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.96 (9.980) | 63.78 (9.470) | 57.37 (19.984)
  CD45+CD3+CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+;D1;1 h;n=1,3,1,5,4,9 | 50.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.66 (4.707) | 67.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.58 (8.122) | 62.71 (13.023) | 55.80 (21.386)
  CD45+CD3+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD69+;D1;6 h;n=1,3,1,5,4,11 | 63.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.49 (3.426) | 80.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.24 (7.910) | 63.26 (12.922) | 60.07 (19.171)
  CD45+CD3+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD69+; D2; n=0,0,1,2,0,1 |  |  | 68.61 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.01 (3.783) |  | 62.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD69+; D8; n=1,3,0,5,4,8 | 58.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 59.29 (5.515) |  | 64.97 (2.165) | 65.73 (6.597) | 51.29 (13.826)
  CD45+CD3+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+; D15;S1; n=1,3,1,5,4,9 | 53.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.92 (4.016) | 72.73 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.08 (6.604) | 58.46 (3.564) | 53.38 (21.988)
  CD45+CD3+CD69+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+; D15;S2; n=0,0,1,0,0,0 |  |  | 67.36 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD69+; D29; n=1,3,1,4,4,8 | 60.54 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.97 (4.090) | 52.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.52 (6.451) | 63.88 (5.978) | 53.68 (19.308)
  CD45+CD3+CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD69+; FU;n=1,2,0,3,1,4 | 54.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.87 (8.259) |  | 68.45 (0.841) | 64.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.21 (17.378)
  CD45+CD3+CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+; USC;n=0,0,1,0,0,0 |  |  | 42.30 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD107+;D1pre; n=1,3,1,5,4,9 | 3.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.70 (6.236) | 11.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.13 (10.732) | 8.92 (4.982) | 8.99 (4.894)
  CD45+CD3+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD107+;D1;1 h;n=1,3,1,5,4,9 | 3.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.63 (8.846) | 1.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.84 (10.971) | 6.79 (3.717) | 7.91 (4.880)
  CD45+CD3+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD107+;D1;6 h;n=1,3,1,5,4,11 | 5.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.98 (6.511) | 24.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.53 (10.804) | 7.25 (3.529) | 11.04 (4.474)
  CD45+CD3+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD107+; D2; n=0,0,1,2,0,1 |  |  | 15.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.17 (2.397) |  | 9.61 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD107+; D8; n=1,3,0,5,4,8 | 19.48 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.93 (4.733) |  | 12.31 (7.851) | 9.81 (6.276) | 10.61 (7.576)
  CD45+CD3+CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD107+; D15;S1; n=1,3,1,5,4,9 | 10.68 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.32 (2.680) | 76.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.84 (7.608) | 8.13 (4.504) | 10.75 (6.692)
  CD45+CD3+CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 84.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD107+; D29; n=1,3,1,4,4,8 | 11.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.24 (3.455) | 54.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.88 (12.246) | 10.30 (6.320) | 10.79 (4.881)
  CD45+CD3+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD107+; FU;n=1,2,0,3,1,4 | 6.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.19 (6.124) |  | 27.28 (11.058) | 5.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.44 (10.953)
  CD45+CD3+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD107+; USC;n=0,0,1,0,0,0 |  |  | 11.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107+;D1pre; n=1,3,1,5,4,9 | 3.22 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 13.33 (5.965) | 11.31 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.68 (10.738) | 8.62 (4.781) | 8.55 (4.996)
  CD45+CD3+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107+;D1;1 h;n=1,3,1,5,4,9 | 3.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.15 (8.408) | 1.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.33 (10.922) | 6.42 (3.287) | 7.43 (4.929)
  CD45+CD3+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 5.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.29 (5.756) | 24.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.00 (10.573) | 6.89 (3.217) | 10.03 (4.618)
  CD45+CD3+CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 15.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 6.02 (2.220) |  | 9.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD69+CD107+; D8; n=1,3,0,5,4,8 | 17.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.29 (3.881) |  | 11.95 (7.603) | 9.36 (5.904) | 9.58 (6.752)
  CD45+CD3+CD69+CD107+; D15;S1 ; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107+; D15;S1 ; n=1,3,1,5,4,9 | 9.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.25 (2.622) | 62.5 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.63 (7.568) | 7.74 (4.077) | 10.13 (6.879)
  CD45+CD3+CD69+CD107+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+CD107+; D15; S2; n=0,0,1,0,0,0 |  |  | 61.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD69+CD107+; D29; n=1,3,1,4,4,8 | 10.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.07 (3.421) | 40.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.47 (11.821) | 9.88 (5.888) | 9.56 (4.499)
  CD45+CD3+CD69+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD69+CD107+; FU;n=1,2,0,3,1,4 | 5.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.98 (5.961) |  | 26.15 (10.446) | 4.98 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.70 (9.912)
  CD45+CD3+CD69+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+CD107+; USC;n=0,0,1,0,0,0 |  |  | 10.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107-;D1pre; n=1,3,1,5,4,9 | 46.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 51.06 (3.578) | 50.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.28 (8.029) | 55.15 (13.699) | 48.82 (16.871)
  CD45+CD3+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107-;D1;1 h;n=1,3,1,5,4,9 | 47.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 48.51 (4.092) | 65.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 51.25 (7.800) | 56.29 (13.709) | 48.37 (18.392)
  CD45+CD3+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 57.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.20 (6.989) | 55.50 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.24 (5.794) | 56.37 (14.071) | 50.04 (16.622)
  CD45+CD3+CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 53.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.99 (6.003) |  | 53.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD69+CD107-; D8; n=1,3,0,5,4,8 | 40.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.00 (5.550) |  | 53.02 (7.641) | 56.37 (8.661) | 41.72 (11.909)
  CD45+CD3+CD69+CD107-; D15; S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69+CD107-; D15; S1; n=1,3,1,5,4,9 | 44.09 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.67 (5.732) | 10.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.45 (4.502) | 50.72 (6.589) | 43.25 (18.831)
  CD45+CD3+CD69+CD107-; D15; S2;n=0, 0, 1, 0, 0, 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+CD107-; D15; S2;n=0, 0, 1, 0, 0, 0 |  |  | 6.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD69+CD107-; D29; n=1,3,1,4,4,8 | 50.26 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 58.89 (0.756) | 12.29 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.05 (6.415) | 54.00 (11.624) | 44.11 (17.898)
  CD45+CD3+CD69+CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD69+CD107-; FU;n=1,2,0,3,1,4 | 48.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 57.90 (2.298) |  | 42.29 (9.606) | 59.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 55.52 (16.825)
  CD45+CD3+CD69+CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69+CD107-; USC;n=0,0,1,0,0,0 |  |  | 31.83 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69-CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107+;D1pre; n=1,3,1,5,4,9 | 0.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.36 (0.277) | 0.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.45 (0.579) | 0.30 (0.324) | 0.44 (0.537)
  CD45+CD3+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107+;D1;1 h;n=1,3,1,5,4,9 | 0.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.47 (0.451) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.50 (0.615) | 0.36 (0.477) | 0.48 (0.459)
  CD45+CD3+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.69 (0.777) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.54 (0.844) | 0.36 (0.349) | 1.01 (1.233)
  CD45+CD3+CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.15 (0.177) |  | 0.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD69-CD107+; D8; n=1,3,0,5,4,8 | 1.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.64 (0.861) |  | 0.35 (3.392) | 0.45 (0.458) | 1.04 (1.201)
  CD45+CD3+CD69-CD107+; D15; S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107+; D15; S1; n=1,3,1,5,4,9 | 0.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.07 (0.059) | 13.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.21 (0.187) | 0.39 (0.439) | 0.62 (0.460)
  CD45+CD3+CD69-CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69-CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 23.43 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD69-CD107+; D29; n=1,3,1,4,4,8 | 1.34 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.17 (0.042) | 13.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.41 (0.476) | 0.42 (0.449) | 1.22 (1.608)
  CD45+CD3+CD69-CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD69-CD107+; FU;n=1,2,0,3,1,4 | 0.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.23 (0.163) |  | 1.13 (0.705) | 0.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.75 (1.090)
  CD45+CD3+CD69-CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69-CD107+; USC;n=0,0,1,0,0,0 |  |  | 1.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69-CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107-;D1pre; n=1,3,1,5,4,9 | 50.23 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.23 (2.664) | 37.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 34.58 (9.638) | 35.93 (9.242) | 42.20 (19.537)
  CD45+CD3+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107-;D1;1 h;n=1,3,1,5,4,9 | 49.71 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 38.87 (5.156) | 32.84 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.91 (7.854) | 36.93 (12.789) | 43.72 (21.074)
  CD45+CD3+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 36.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 37.83 (3.625) | 20.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 37.23 (7.810) | 36.38 (12.700) | 38.92 (18.214)
  CD45+CD3+CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 31.39 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 30.85 (3.606) |  | 37.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD69-CD107-; D8; n=1,3,0,5,4,8 | 40.39 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 40.07 (5.758) |  | 34.67 (2.320) | 33.83 (6.576) | 47.67 (13.646)
  CD45+CD3+CD69-CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD69-CD107-; D15;S1; n=1,3,1,5,4,9 | 45.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.01 (3.981) | 13.64 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 34.71 (6.524) | 41.15 (3.409) | 46.00 (21.556)
  CD45+CD3+CD69-CD107-; D15; S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69-CD107-; D15; S2;n=0,0,1,0,0,0 |  |  | 9.2 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD69-CD107-; D29; n=1,3,1,4,4,8 | 38.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 31.87 (4.127) | 33.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 38.07 (6.801) | 35.70 (5.601) | 45.10 (18.361)
  CD45+CD3+CD69-CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD69-CD107-; FU;n=1,2,0,3,1,4 | 45.14 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 30.91 (8.422) |  | 30.43 (1.483) | 34.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 32.05 (17.570)
  CD45+CD3+CD69-CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD69-CD107-; USC;n=0,0,1,0,0,0 |  |  | 56.55 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+;D1pre; n=1,3,1,5,4,9 | 47.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.18 (3.198) | 63.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.39 (9.372) | 58.78 (9.546) | 52.12 (20.035)
  CD45+CD3+CD8-CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+;D1;1 h;n=1,3,1,5,4,9 | 49.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 58.34 (5.829) | 67.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.93 (7.196) | 59.04 (12.906) | 51.86 (22.844)
  CD45+CD3+CD8-CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD69+;D1;6 h;n=1,3,1,5,4,11 | 62.61 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.24 (3.832) | 77.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 58.97 (6.452) | 59.18 (13.744) | 56.19 (18.029)
  CD45+CD3+CD8-CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD69+; D2; n=0,0,1,2,0,1 |  |  | 67.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 63.36 (5.169) |  | 51.49 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD69+; D8; n=1,3,0,5,4,8 | 57.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 56.36 (7.227) |  | 61.41 (3.385) | 64.59 (10.317) | 42.80 (13.006)
  CD45+CD3+CD8-CD69+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+; D15; S1;n=1,3,1,5,4,9 | 47.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.16 (6.272) | 75.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 61.57 (4.769) | 53.99 (7.004) | 49.92 (22.128)
  CD45+CD3+CD8-CD69+; D15; S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+; D15; S2;n=0,0,1,0,0,0 |  |  | 66.87 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD69+; D29; n=1,3,1,4,4,8 | 59.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 66.23 (5.538) | 54.82 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 57.72 (3.694) | 59.41 (7.751) | 50.71 (19.479)
  CD45+CD3+CD8-CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD69+; FU;n=1,2,0,3,1,4 | 52.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 65.54 (8.811) |  | 62.68 (3.581) | 64.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 59.43 (17.448)
  CD45+CD3+CD8-CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+; USC;n=0,0,1,0,0,0 |  |  | 41.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD107+;D1pre; n=1,3,1,5,4,9 | 1.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.52 (6.264) | 8.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.13 (7.030) | 9.40 (9.095) | 8.89 (7.406)
  CD45+CD3+CD8-CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD107+;D1;1 h;n=1,3,1,5,4,9 | 2.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.13 (9.350) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.77 (6.304) | 10.14 (11.064) | 5.52 (3.023)
  CD45+CD3+CD8-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD107+;D1;6 h;n=1,3,1,5,4,11 | 4.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.43 (6.165) | 14.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.25 (7.708) | 11.10 (12.927) | 8.49 (3.930)
  CD45+CD3+CD8-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD107+; D2; n=0,0,1,2,0,1 |  |  | 7.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 22.06 (12.183) |  | 12.25 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD107+; D8; n=1,3,0,5,4,8 | 16.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.43 (4.942) |  | 8.44 (5.762) | 6.89 (3.550) | 7.20 (3.406)
  CD45+CD3+CD8-CD107+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD107+; D15; S1;n=1,3,1,5,4,9 | 8.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.31 (2.868) | 67.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.32 (4.700) | 6.66 (4.113) | 10.03 (7.687)
  CD45+CD3+CD8-CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 79.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD107+; D29; n=1,3,1,4,4,8 | 6.04 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.33 (3.967) | 45.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.99 (2.600) | 8.29 (3.475) | 8.07 (5.728)
  CD45+CD3+CD8-CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD107+; FU;n=1,2,0,3,1,4 | 3.99 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 12.22 (14.015) |  | 16.79 (8.978) | 4.78 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 16.10 (11.466)
  CD45+CD3+CD8-CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD107+; USC;n=0,0,1,0,0,0 |  |  | 10.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107+;D1pre; n=1,3,1,5,4,9 | 1.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.34 (6.086) | 8.62 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.66 (6.705) | 8.70 (8.036) | 8.49 (7.511)
  CD45+CD3+CD8-CD69+CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107+;D1;1 h;n=1,3,1,5,4,9 | 2.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.84 (8.957) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 8.39 (6.132) | 9.37 (9.954) | 5.08 (3.208)
  CD45+CD3+CD8-CD69+CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD69+CD107+;D1;6 h;n=1,3,1,5,4,11 | 4.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.99 (5.509) | 14.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 9.81 (7.518) | 10.26 (11.433) | 7.64 (3.879)
  CD45+CD3+CD8-CD69+CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD69+CD107+; D2; n=0,0,1,2,0,1 |  |  | 7.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 20.45 (10.684) |  | 11.90 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD69+CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD69+CD107+; D8; n=1,3,0,5,4,8 | 15.40 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.16 (4.542) |  | 8.22 (5.569) | 6.68 (3.439) | 6.35 (3.062)
  CD45+CD3+CD8-CD69+CD107+; D15; S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107+; D15; S1;n=1,3,1,5,4,9 | 7.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 4.28 (2.851) | 62.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.09 (4.543) | 6.42 (3.978) | 9.27 (7.216)
  CD45+CD3+CD8-CD69+CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 58.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD69+CD107+; D29; n=1,3,1,4,4,8 | 5.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 5.26 (3.913) | 38.58 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 7.39 (1.938) | 8.03 (3.389) | 6.92 (4.718)
  CD45+CD3+CD8-CD69+CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD69+CD107+; FU;n=1,2,0,3,1,4 | 3.94 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 11.93 (13.598) |  | 16.09 (8.306) | 4.63 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 14.87 (10.444)
  CD45+CD3+CD8-CD69+CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+CD107+; USC;n=0,0,1,0,0,0 |  |  | 9.71 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107-;D1pre; n=1,3,1,5,4,9 | 46.02 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.84 (2.952) | 55.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 51.72 (7.637) | 50.08 (9.719) | 43.63 (15.780)
  CD45+CD3+CD8-CD69+CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107-;D1;1 h;n=1,3,1,5,4,9 | 47.12 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 49.48 (3.288) | 67.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.53 (6.408) | 49.68 (9.756) | 46.78 (20.420)
  CD45+CD3+CD8-CD69+CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD69+CD107-;D1;6 h;n=1,3,1,5,4,11 | 57.92 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 52.25 (6.443) | 62.93 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 49.16 (4.649) | 48.93 (11.819) | 48.55 (16.115)
  CD45+CD3+CD8-CD69+CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD69+CD107-; D2; n=0,0,1,2,0,1 |  |  | 59.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 42.91 (5.515) |  | 39.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD69+CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD69+CD107-; D8; n=1,3,0,5,4,8 | 41.88 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 51.21 (6.451) |  | 53.19 (5.196) | 57.91 (9.965) | 36.45 (12.237)
  CD45+CD3+CD8-CD69+CD107-; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69+CD107-; D15;S1; n=1,3,1,5,4,9 | 40.25 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 59.88 (3.546) | 13.79 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 54.48 (6.572) | 47.58 (6.986) | 40.65 (18.749)
  CD45+CD3+CD8-CD69+CD107-; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+CD107-; D15;S2; n=0,0,1,0,0,0 |  |  | 8.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69+CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD69+CD107-; D29; n=1,3,1,4,4,8 | 53.36 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 60.98 (1.681) | 16.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 50.33 (5.623) | 51.37 (5.812) | 43.79 (19.299)
  CD45+CD3+CD8-CD69+CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD69+CD107-; FU;n=1,2,0,3,1,4 | 48.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 53.62 (4.794) |  | 46.59 (4.968) | 60.09 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 44.55 (12.109)
  CD45+CD3+CD8-CD69+CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69+CD107-; USC;n=0,0,1,0,0,0 |  |  | 31.33 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69-CD107+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107+;D1pre; n=1,3,1,5,4,9 | 0.01 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.17 (0.180) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.47 (0.607) | 0.70 (1.089) | 0.41 (0.541)
  CD45+CD3+CD8-CD69-CD107+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107+;D1;1 h;n=1,3,1,5,4,9 | 0.03 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.27 (0.414) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.38 (0.526) | 0.77 (1.174) | 0.43 (0.496)
  CD45+CD3+CD8-CD69-CD107+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD69-CD107+;D1;6 h;n=1,3,1,5,4,11 | 0.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.44 (0.691) | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.44 (0.695) | 0.85 (1.537) | 0.85 (1.277)
  CD45+CD3+CD8-CD69-CD107+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD69-CD107+; D2; n=0,0,1,2,0,1 |  |  | 0.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.62 (1.492) |  | 0.35 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD69-CD107+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD69-CD107+; D8; n=1,3,0,5,4,8 | 1.19 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.27 (0.406) |  | 0.22 (0.239) | 0.21 (0.194) | 0.85 (0.855)
  CD45+CD3+CD8-CD69-CD107+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107+; D15;S1; n=1,3,1,5,4,9 | 0.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.02 (0.020) | 5.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.23 (0.217) | 0.25 (0.179) | 0.76 (0.966)
  CD45+CD3+CD8-CD69-CD107+; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69-CD107+; D15;S2; n=0,0,1,0,0,0 |  |  | 21.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69-CD107+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD69-CD107+; D29; n=1,3,1,4,4,8 | 0.24 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.08 (0.057) | 7.11 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.60 (0.787) | 0.23 (0.117) | 1.15 (1.764)
  CD45+CD3+CD8-CD69-CD107+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD69-CD107+; FU;n=1,2,0,3,1,4 | 0.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 0.30 (0.417) |  | 0.70 (0.729) | 0.15 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 1.22 (1.319)
  CD45+CD3+CD8-CD69-CD107+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69-CD107+; USC;n=0,0,1,0,0,0 |  |  | 0.91 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69-CD107-;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107-;D1pre; n=1,3,1,5,4,9 | 52.08 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 38.64 (3.370) | 36.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 39.14 (9.186) | 40.53 (9.843) | 47.48 (19.639)
  CD45+CD3+CD8-CD69-CD107-;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107-;D1;1 h;n=1,3,1,5,4,9 | 50.83 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 41.39 (6.239) | 32.81 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 38.69 (6.983) | 40.19 (13.401) | 47.70 (22.541)
  CD45+CD3+CD8-CD69-CD107-;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3+CD8-CD69-CD107-;D1;6 h;n=1,3,1,5,4,11 | 37.28 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 39.32 (4.165) | 22.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 40.59 (6.401) | 39.98 (14.362) | 42.96 (17.217)
  CD45+CD3+CD8-CD69-CD107-; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3+CD8-CD69-CD107-; D2; n=0,0,1,2,0,1 |  |  | 32.89 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.03 (6.661) |  | 48.16 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3+CD8-CD69-CD107-; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3+CD8-CD69-CD107-; D8; n=1,3,0,5,4,8 | 41.53 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 43.36 (7.367) |  | 38.37 (3.532) | 35.20 (10.279) | 56.36 (12.433)
  CD45+CD3+CD8-CD69-CD107-; D15;S1;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3+CD8-CD69-CD107-; D15;S1;n=1,3,1,5,4,9 | 51.72 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 35.82 (6.285) | 18.97 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 38.20 (4.657) | 45.76 (6.941) | 49.32 (21.812)
  CD45+CD3+CD8-CD69-CD107-; D15;S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69-CD107-; D15;S2; n=0,0,1,0,0,0 |  |  | 11.4 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3+CD8-CD69-CD107-; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3+CD8-CD69-CD107-; D29; n=1,3,1,4,4,8 | 40.59 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 33.69 (5.590) | 38.07 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 41.69 (3.048) | 40.37 (7.766) | 48.14 (18.661)
  CD45+CD3+CD8-CD69-CD107-; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3+CD8-CD69-CD107-; FU;n=1,2,0,3,1,4 | 47.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 34.17 (9.228) |  | 36.61 (4.300) | 35.13 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 39.35 (17.631)
  CD45+CD3+CD8-CD69-CD107-; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3+CD8-CD69-CD107-; USC;n=0,0,1,0,0,0 |  |  | 58.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD19+CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+CD69+;D1pre; n=1,3,1,5,4,9 | 75.76 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 67.04 (8.518) | 84.75 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.41 (7.715) | 66.51 (16.098) | 60.06 (14.370)
  CD45+CD3-CD19+CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+CD69+;D1;1 h;n=1,3,1,5,4,9 | 80.05 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 66.03 (12.856) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.80 (9.542) | 67.42 (15.190) | 61.79 (14.941)
  CD45+CD3-CD19+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD3-CD19+CD69+;D1;6 h;n=1,3,1,5,4,11 | 78.69 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 69.97 (8.412) | 84.21 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.55 (5.810) | 63.22 (18.089) | 66.22 (20.094)
  CD45+CD3-CD19+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD3-CD19+CD69+; D2; n=0,0,1,2,0,1 |  |  | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 71.53 (0.721) |  | 58.57 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD3-CD19+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD3-CD19+CD69+; D8; n=1,3,0,5,4,8 | 72.44 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 62.85 (5.952) |  | 70.60 (5.653) | 66.95 (20.328) | 52.90 (52.90)
  CD45+CD3-CD19+CD69+; D15;S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD3-CD19+CD69+; D15;S1; n=1,3,1,5,4,9 | 71.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 64.28 (7.449) | 89.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.07 (6.942) | 61.50 (12.596) | 61.77 (61.77)
  CD45+CD3-CD19+CD69+; D15;S2;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD19+CD69+; D15;S2;n=0,0,1,0,0,0 |  |  | 85.95 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD3-CD19+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD3-CD19+CD69+; D29; n=1,3,1,4,4,8 | 74.65 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 72.22 (17.828) | 66.18 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.83 (5.767) | 65.80 (7.211) | 61.49 (61.49)
  CD45+CD3-CD19+CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD3-CD19+CD69+; FU;n=1,2,0,3,1,4 | 74.67 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 68.44 (5.268) |  | 73.60 (7.363) | 73.22 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 70.54 (70.54)
  CD45+CD3-CD19+CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD3-CD19+CD69+; USC;n=0,0,1,0,0,0 |  |  | 60.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD14+CD69+;D1pre; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+CD69+;D1pre; n=1,3,1,5,4,9 | 99.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.57 (0.371) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.27 (0.308) | 99.19 (1.046) | 99.39 (0.407)
  CD45+CD14+CD69+;D1;1 h;n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+CD69+;D1;1 h;n=1,3,1,5,4,9 | 99.86 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.54 (0.204) | 99.55 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.42 (0.202) | 99.51 (0.658) | 99.37 (0.725)
  CD45+CD14+CD69+;D1;6 h;n=1,3,1,5,4,11: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 11
  CD45+CD14+CD69+;D1;6 h;n=1,3,1,5,4,11 | 99.45 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.19 (0.239) | 99.78 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.28 (0.393) | 99.11 (1.442) | 99.24 (0.942)
  CD45+CD14+CD69+; D2; n=0,0,1,2,0,1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1
  CD45+CD14+CD69+; D2; n=0,0,1,2,0,1 |  |  | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.16 (1.018) |  | 99.06 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point.
  CD45+CD14+CD69+; D8; n=1,3,0,5,4,8: number analyzed (Participants) | 1 | 3 | 0 | 5 | 4 | 8
  CD45+CD14+CD69+; D8; n=1,3,0,5,4,8 | 99.41 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.49 (0.297) |  | 99.15 (0.763) | 99.78 (0.241) | 98.64 (1.993)
  CD45+CD14+CD69+; D15; S1; n=1,3,1,5,4,9: number analyzed (Participants) | 1 | 3 | 1 | 5 | 4 | 9
  CD45+CD14+CD69+; D15; S1; n=1,3,1,5,4,9 | 99.37 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.70 (0.145) | 100.00 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.71 (0.311) | 99.50 (0.435) | 97.67 (3.444)
  CD45+CD14+CD69+; D15; S2; n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD14+CD69+; D15; S2; n=0,0,1,0,0,0 |  |  | 99.74 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |
  CD45+CD14+CD69+; D29; n=1,3,1,4,4,8: number analyzed (Participants) | 1 | 3 | 1 | 4 | 4 | 8
  CD45+CD14+CD69+; D29; n=1,3,1,4,4,8 | 99.66 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.61 (0.391) | 98.85 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.53 (0.379) | 99.68 (0.225) | 98.98 (1.950)
  CD45+CD14+CD69+; FU;n=1,2,0,3,1,4: number analyzed (Participants) | 1 | 2 | 0 | 3 | 1 | 4
  CD45+CD14+CD69+; FU;n=1,2,0,3,1,4 | 99.71 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.66 (0.028) |  | 99.62 (0.219) | 99.47 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 99.65 (0.288)
  CD45+CD14+CD69+; USC;n=0,0,1,0,0,0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  CD45+CD14+CD69+; USC;n=0,0,1,0,0,0 |  |  | 96.17 (NA) — Standard deviation could not be calculated as a single participant was analyzed at the specified time point. |  |  |

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of study treatment until 45 days or 5 half-lives from the last dose of study treatment (median of 6.143 weeks of drug exposure).
Description: AEs and SAEs were collected in the All Treated Population which comprised of all participants who received at least one dose of GSK2849330. Treatment groups with same dose and administration frequency were combined as pre-specified in reporting and analysis plan.
Arm/Group | GSK2849330 1.4 mg/kg Weekly | GSK2849330 3 mg/kg Every 2 Weeks | GSK2849330 3 mg/kg Weekly | GSK2849330 10 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Every 2 Weeks | GSK2849330 30 mg/kg Weekly
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/2 | 0/5 | 0/4 | 1/14
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 0/2 | 1/5 | 1/4 | 3/14
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2 | 5/5 | 4/4 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2849330 1.4 mg/kg Weekly (N=1) | GSK2849330 3 mg/kg Every 2 Weeks (N=3) | GSK2849330 3 mg/kg Weekly (N=2) | GSK2849330 10 mg/kg Every 2 Weeks (N=5) | GSK2849330 30 mg/kg Every 2 Weeks (N=4) | GSK2849330 30 mg/kg Weekly (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2849330 1.4 mg/kg Weekly (N=1) | GSK2849330 3 mg/kg Every 2 Weeks (N=3) | GSK2849330 3 mg/kg Weekly (N=2) | GSK2849330 10 mg/kg Every 2 Weeks (N=5) | GSK2849330 30 mg/kg Every 2 Weeks (N=4) | GSK2849330 30 mg/kg Weekly (N=14)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (3) | 2 (2) | 3 (4) | 9 (12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 10 (12)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Cough (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-01-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT01966445/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT01966445/SAP_001.pdf